

#### Protocol for Study M16-560

Rheumatoid Arthritis: Antibody Drug Conjugate ABBV-3373 Vs Adalimumab in Subjects with Moderate to Severe Rheumatoid Arthritis

VERSION: 5.0 DATE: 04 September 2020

SPONSOR: For Non-EU Countries:\* NUMBER OF 40

AbbVie SITES:

1 North Waukegan Road

Bldg. AP31

North Chicago, IL 60064

USA

For EU Countries:\*
AbbVie Deutschland
GmbH & Co. KG (AbbVie)

Knollstrasse 50 67061 Ludwigshafen

Germany

ABBVIE INVESTIGATIONAL ABBV-3373 EUDRACT: 2018-003053-21

PRODUCT:

FULL TITLE: A Randomized, Double-Blind, Double-Dummy, Active Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABBV-3373 in Subjects with Moderate to Severe Rheumatoid Arthritis

Incorporating Versions 1.0, 2.0, 3.0, 4.0, and 5.0

PRINCIPAL INVESTIGATOR(S): Investigator information on file at AbbVie.

SPONSOR/EMERGENCY MEDICAL

CONTACT:\*

AbbVie Deutschland GmbH & Co. KG

Knollstrasse

67061 Ludwigshafen

Germany

Office:
Mobile:
Fax:
Email:

EMERGENCY 24 hour Number: +1 973-784-6402

<sup>\*</sup>The specific contact details of the AbbVie legal/regulatory entity (person) within the relevant country are provided within the clinical trial agreement with the Investigator/Institution and in the Clinical Trial Application with the Competent Authority. Additional study contact information can be found in the Operations Manual (Appendix L).



# **TABLE OF CONTENTS**

| <u>1</u> | SYNOPSIS | 5 |
|----------|-----------------------------------------------------|----|
| <u>2</u> | INTRODUCTION | 8 |
| 2.1 | BACKGROUND AND RATIONALE | 8 |
| 2.2 | BENEFITS AND RISKS TO SUBJECTS | 8 |
| <u>3</u> | STUDY OBJECTIVES AND ENDPOINTS | 9 |
| 3.1 | OBJECTIVES | 9 |
| 3.2 | PRIMARY ENDPOINT | 10 |
| 3.3 | SECONDARY AND ADDITIONAL ENDPOINTS | 10 |
| 3.4 | SAFETY ENDPOINTS | 10 |
| 3.5 | PHARMACOKINETIC AND IMMUNOGENICITY ENDPOINTS | 11 |
| 3.6 | 5 BIOMARKER ENDPOINTS | 11 |
| <u>4</u> | INVESTIGATIONAL PLAN | 11 |
| 4.1 | OVERALL STUDY DESIGN AND PLAN | 11 |
| 4.2 | 2 DISCUSSION OF STUDY DESIGN | 13 |
| <u>5</u> | STUDY ACTIVITIES | 14 |
| 5.1 | L ELIGIBILITY CRITERIA | 14 |
| 5.2 | 2 CONTRACEPTION RECOMMENDATIONS | 17 |
| 5.3 | PROHIBITED MEDICATIONS AND THERAPY | 18 |
| 5.4 | PRIOR AND CONCOMITANT THERAPY | 18 |
| 5.5 | WITHDRAWAL OF SUBJECTS AND DISCONTINUATION OF STUDY | 19 |
| 5.6 | FOLLOW-UP FOR SUBJECT WITHDRAWAL FROM STUDY | 20 |
| 5.7 | STUDY DRUG | 21 |
| 5.8 | RANDOMIZATION/DRUG ASSIGNMENT | 22 |
| 5.9 | PROTOCOL DEVIATIONS | 23 |
| <u>6</u> | SAFETY CONSIDERATIONS | 23 |
| 6.1 | COMPLAINTS AND ADVERSE EVENTS | 23 |
| 6.2 | 2 TOXICITY MANAGEMENT | 27 |



| <u>7</u> | STATISTICAL METHODS & DETERMINATION OF SAMPLE SIZE | 30 |
|---|---|---|
| 7.1 | STATISTICAL AND ANALYTICAL PLANS | 30 |
| 7.2 | DEFINITION FOR ANALYSIS POPULATIONS | 30 |
| 7.3 | STATISTICAL ANALYSES FOR EFFICACY | 31 |
| 7.4 | STATISTICAL ANALYSES FOR SAFETY | 33 |
| 7.5 | STATISTICAL ANALYSIS OF PHARMACOKINETIC AND IMMUNOGENITICY DATA | 33 |
| 7.6 | STATISTICAL ANALYSIS OF BIOMARKER DATA | 33 |
| 7.7 | Interim Analysis | 33 |
| <u>8</u> | ETHICS | 34 |
| 8.1 | INDEPENDENT ETHICS COMMITTEE/INSTITUTIONAL REVIEW BOARD (IEC/IRB) | 34 |
| 8.2 | ETHICAL CONDUCT OF THE STUDY | 34 |
| 8.3 | Subject Confidentiality | 34 |
| <u>9</u> | SOURCE DOCUMENTS AND CASE REPORT FORM COMPLETION | 34 |
| <u>10</u> | DATA QUALITY ASSURANCE | 34 |
| <u>11</u> | COMPLETION OF THE STUDY | 35 |
| <u>12</u> | REFERENCES | 35 |
| LIS | T OF TABLES | |
| TAE | BLE 1. IDENTITY OF INVESTIGATIONAL PRODUCT | 22 |
| TAE | SLE 2. SPECIFIC TOXICITY MANAGEMENT GUIDELINES FOR ABNORMAL LABORATORY VALUES | 28 |
| LIS | T OF FIGURES | |
| FIG | URE 1. STUDY SCHEMATIC | 12 |
| LIS | T OF APPENDICES | |
| APF | PENDIX A. STUDY SPECIFIC ABBREVIATIONS AND TERMS | 36 |
| APF | PENDIX B. RESPONSIBILITIES OF THE INVESTIGATOR | 39 |



| APPENDIX C. | LIST OF PROTOCOL SIGNATORIES | 40 |
|-------------|--------------------------------------------------|----|
| APPENDIX D. | ADDITIONAL ENDPOINT/ASSESSMENT DEFINITIONS | 41 |
| APPENDIX E. | JOINT EVALUATION WORKSHEET EXAMPLE | 43 |
| APPENDIX F. | REPORTED OUTCOMES VAS | 44 |
| APPENDIX G. | HEALTH ASSESSMENT QUESTIONNAIRE DISABILITY INDEX | 45 |
| APPENDIX H. | 36-ITEM SHORT FORM HEALTH SURVEY SAMPLE | 46 |
| APPENDIX I. | RHEUMATOLOGY COMMON TOXICITY CRITERIA V.2.0 | 47 |
| APPENDIX J. | ACTIVITY SCHEDULE | 61 |
| APPENDIX K. | SUMMARY OF CHANGES | 65 |
| APPENDIX L. | OPERATIONS MANUAL | 68 |



#### 1 SYNOPSIS

Title: A Randomized, Double-Blind, Double-Dummy, Active Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABBV-3373 in Subjects with Moderate to Severe Rheumatoid Arthritis

#### **Background and Rationale:**

Tumor necrosis factor (TNF) $\alpha$  antagonists are considered effective therapies with established safety profiles in patients with immune-mediated inflammatory diseases, including rheumatoid arthritis (RA). Nevertheless, TNF $\alpha$  antagonists as well as other biologics and targeted synthetic disease-modifying antirheumatic drugs (DMARDs) provide 50% improvement in arthritis scores (ACR50) for fewer than half of RA subjects, even in combination with methotrexate (MTX), indicating that there remains an unmet clinical need for improved therapies.

Glucocorticoid receptor modulators (GRMs) are potent drugs for treating many inflammatory diseases, including RA. However, the full efficacy of GRM therapy is not achieved with existing agents due to systemic side effects.

ABBV-3373 is an antibody-drug conjugate (ADC) composed of adalimumab (the active component of Humira®) conjugated to A-1677770, a proprietary, highly potent GRM (also referred to as the payload) being developed for the treatment of immune-mediated inflammatory diseases including RA. This adalimumab/GRM ADC has the potential to deliver a highly potent anti-inflammatory payload selectively to the activated immune cells that express transmembrane TNF, and meanwhile to minimize systemic exposure to the free payload GRM. Therefore, the adalimumab/GRM ADC is a promising novel therapeutic agent which can achieve transformational efficacy relative to adalimumab while reducing side effects caused by free GRM systemic exposure.

#### Objective(s) and Endpoint(s):

#### Primary

- To assess the safety, tolerability, and efficacy of ABBV-3373
   administered every other week (eow) intravenously (IV) in
   subjects with moderately to severely active RA on background
   MTX.
- To compare clinical efficacy of ABBV-3373 with adalimumab and to test the concept that an anti-TNF antibody-drug-conjugate has the potential to provide superior efficacy than the traditional anti-TNF antibody in RA.

#### Secondary

- To compare adalimumab with synthetic placebo control to establish assay sensitivity.
- To assess the pharmacokinetics (PK), pharmacodynamics and immunogenicity of ABBV-3373.
- To assess the durability of the treatment effect of ABBV-3373 after discontinuation.



| | Primary Endpoint: The change in disease activity score (DAS)28 (C-reactive protein [CRP]) from Baseline (BL) at Week 12. |
|---|---|
| Investigator(s): | Multi-center. |
| Study Site(s): | Approximately 40 sites; United States, Puerto Rico, Germany, Hungary, Israel, Netherlands, Poland. |
| Study Population and Number of<br>Subjects to be Enrolled: | The study population consists of adults with moderate to severe RA. Approximately 45 subjects will be enrolled. |
| Investigational Plan: | This is a randomized, double-blind, double-dummy, adalimumab active-controlled (12-week) Phase 2a study to assess the safety, tolerability, PK, pharmacodynamics, immunogenicity and efficacy following multiple IV administrations of ABBV-3373 or multiple subcutaneous (SC) injections of adalimumab in subjects with RA on background MTX. In the actively controlled period of the first 12 weeks of treatment, 45 subjects will receive either ABBV-3373 100 mg IV and the matching placebo for adalimumab SC eow or in the control arm the matching placebo for ABBV-3373 IV and adalimumab 80 mg SC eow (double-dummy) according to a 2:1 ratio. Thereafter, all subjects enter a 12-week double-blind extension period. At Week 12, the administration of ABBV-3373 will stop (i.e., the last dose of ABBV-3373 will be given at Week 10) to assess the durability of the observed clinical effects up to 24 weeks. To keep blinding of the study beyond Week 12, the subjects randomized to ABBV-3373 will receive placebo injections, whereas subjects randomized into the adalimumab arm will continue their 80 mg dosing until Week 22. At Week 12 and within the blinded extension period subjects who have not achieved at least a 20% improvement in both their swollen joint count and tender joint count based on 28 joint assessment compared with BL may be discontinued from the study at the discretion of the Investigator. Subsequently, standard of care may be administered at the discretion of the Investigator. After all endpoints are assessed at Week 24, a telephone contact is planned to follow up on safety 70 days after the last dose. |
| Key Eligibility Criteria: | <ul> <li>Subjects or their legally authorized representative must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.</li> <li>Adult male or female, between 18 and 75 years of age inclusive at Screening.</li> <li>Diagnosis of RA for &gt; 3 months based on the 1987 ACR classification criteria or 2010 ACR/European League against Rheumatism (EULAR) criteria.</li> <li>Subject meets the following disease activity criteria: &gt; 4 swollen joints (based on 28 joint count) and &gt; 4 tender</li> </ul> |
| | ≥ 4 swollen joints (based on 28 joint count) and ≥ 4 tender joints (based on 28 joint count) at Screening and BL Visits; and DAS28(CRP) ≥ 3.2 at Screening. |



| | <ul> <li>Incomplete response to MTX. Subjects must have been on<br/>oral or parenteral MTX therapy ≥ 3 months and on a stable<br/>prescription of 15 to 25 mg/week (or ≥ 10 mg/week in subjects<br/>intolerant of MTX at doses ≥ 15 mg/week) for ≥ 4 weeks prior<br/>to the first dose of study drug. Subject must be expected to<br/>be able to continue on stable dose of MTX for the duration of<br/>study participation.</li> </ul> |
|---|---|
| Study Drug and Duration of Treatment: | ABBV-3373 (50 mg/mL) and matching placebo, adalimumab (80 mg/0.8 mL) and matching placebo. In the first 12 weeks of treatment, subjects will receive either ABBV-3373 100 mg IV and the matching placebo for adalimumab SC eow or in the control arm the matching placebo for ABBV-3373 IV and adalimumab 80 mg SC eow. At Week 12, the administration of ABBV-3373 will stop (i.e., the last dose of ABBV-3373 will be given at Week 10) to assess the durability of the observed clinical effects up to 24 weeks. |
| Date of Protocol Synopsis: | 04 September 2020 |



#### 2 INTRODUCTION

# 2.1 Background and Rationale

#### Why Is This Study Being Conducted

Tumor necrosis factor (TNF) $\alpha$  antagonists reduce the signs and symptoms of disease by reducing inflammation and limiting the progression of tissue destruction and are considered effective therapies with established safety profiles in patients with immune-mediated inflammatory diseases, including rheumatoid arthritis (RA). Nevertheless, TNF $\alpha$  antagonists as well as other biologics and targeted synthetic disease-modifying antirheumatic drugs (DMARDs) provide 50% improvement in arthritis scores (American College of Rheumatology 50% improvement criteria [ACR50]) for fewer than half of RA subjects, even in combination with methotrexate (MTX), indicating that there remains an unmet clinical need for improved therapies.

Glucocorticoid receptor modulators (GRMs) are potent drugs for treating many inflammatory diseases. In RA, GRMs such as prednisone are highly effective at reducing inflammation and fatigue as well as relieving pain. However, the administration of GRMs is limited due to their side effect profile including (but not limited to) hypothalamic-pituitary-adrenal (HPA) axis suppression, increased rates of bone fracture due to osteoporosis, hyperglycemia, glaucoma, skin thinning and weight gain.<sup>1</sup> Thus, the full efficacy of GRM therapy is not achieved with existing agents due to systemic side effects.

ABBV-3373 is an antibody-drug conjugate (ADC) composed of adalimumab (the active component of Humira®) conjugated to A-1677770, a proprietary, highly potent GRM (also referred to as the payload) being developed for the treatment of immune-mediated inflammatory diseases including RA. This adalimumab/GRM ADC has the potential to deliver a highly potent anti-inflammatory payload selectively to the activated immune cells that express transmembrane TNF, and meanwhile to minimize systemic exposure to the free payload GRM. Therefore, the adalimumab/GRM ADC is promising as a novel therapeutic agent which can achieve transformational efficacy relative to adalimumab while reducing side effects caused by free GRM systemic exposure.

#### **Clinical Hypothesis**

ABBV-3373 is safe and well-tolerated and provides superior efficacy in subjects with moderately to severely active RA on background MTX compared to adalimumab.

# 2.2 Benefits and Risks to Subjects

The clinical efficacy of TNF inhibitors and GRMs in the treatment of RA is well established. Based on the preclinical data discussed in the ABBV-3373 Investigator's Brochure, ABBV-3373 is expected to demonstrate therapeutic benefit in treatment of RA and other immune-mediated inflammatory diseases with a favorable safety profile. Preclinical toxicology of ABBV-3373 suggests that the potential risks to human subjects receiving ABBV-3373 treatment are consistent with known effects of adalimumab and glucocorticoids (GCs). ABBV-3373 was tested in a Phase 1 single ascending dose (SAD) study in healthy volunteers in which 6 cohorts of subcutaneous (SC) (30, 100, 300 mg) and intravenous (IV) (30, 300, 900 mg) successfully completed dosing.



Medical review of the available safety data from the Phase 1 study did not identify any unexpected risk or trend to the healthy volunteer population. All single doses tested to date have been well tolerated. For further details, please see the-ABBV-3373 Investigator's Brochure.<sup>2</sup>

In clinical settings, TNF antagonists and GCs have been associated with an increased risk of serious infections due to bacterial, mycobacterial, invasive fungal, viral, parasitic, or other opportunistic pathogens. Opportunistic infections have included tuberculosis (TB) and histoplasmosis. Patients will be closely monitored during the clinical study for any signs of infection.

Tumor necrosis factor antagonists have also been associated with an increased risk for malignancy (including lymphoma), hepatitis B virus (HBV) reactivation, worsening or new onset heart failure, and rarely central nervous system demyelinating disease, pancytopenia including aplastic anemia, and lupus-like syndrome.

The risk of hypersensitivity reaction or other post-dose systemic reaction for humans who receive multiple doses of ABBV-3373 is considered a potential risk. During Study M16-560, 1 case of anaphylactic shock was observed following repeated eow IV (over 3 minute bolus injection) administration of ABBV-3373. The event was assessed by the investigator and AbbVie to be reasonably related to study drug. The administration of biologics may lead to such reactions; therefore, patients will be closely monitored during and post drug administrations.

Hypertension is one of the most commonly reported events for GCs in patients, especially with high doses of GCs. Therefore, blood pressure and other vital signs will be monitored during the trial.

Based on the above considerations, the risk to RA patients receiving multiple doses of ABBV-3373 is considered manageable and acceptable. In addition, based on the population and disease being studied and the anticipation that COVID-19 related risks are not expected to differ substantially between study subjects and the broader population of subjects receiving treatment for RA, no change to the benefit/risk balance for subjects in this study is expected.

# 3 STUDY OBJECTIVES AND ENDPOINTS

# 3.1 Objectives

#### **Primary**

- To assess the safety, tolerability, and efficacy of ABBV-3373 administered every other week (eow) intravenously (IV) in subjects with moderately to severely active RA on background MTX.
- 2. To compare clinical efficacy of ABBV-3373 with adalimumab and to test the concept that an anti-TNF antibody-drug-conjugate has the potential to provide superior efficacy than the traditional anti-TNF antibody in RA.

#### Secondary

- To compare adalimumab with synthetic placebo control to establish assay sensitivity.
- 4. To assess the pharmacokinetics (PK), pharmacodynamics, and immunogenicity of ABBV-3373.
- 5. To assess the duration of the treatment effect of ABBV-3373 after discontinuation.



# 3.2 Primary Endpoint

The primary endpoint is the change in disease activity score (DAS)28 (C-reactive protein [CRP]) from Baseline (BL) at Week 12.

# 3.3 Secondary and Additional Endpoints

#### **Secondary Endpoints**

- 1. Change in clinical disease activity index (CDAI) from BL at Week 12
- 2. Change in simplified disease activity index (SDAI) from BL at Week 12
- 3. Change in disease activity score (28 joints) (DAS28) erythrocyte sedimentation rate (ESR) from BL at Week 12
- Achievement of low disease activity (LDA) (DAS28 [CRP] ≤3.2) at Week 12
- 5. Achievement of American College of Rheumatology (ACR) 50 at Week 12

#### **Additional Endpoints**

- 1. Change from BL in DAS28 (CRP) and DAS28 (ESR) at all visits
- 2. Change from BL in CDAI at all visits
- 3. Change from BL in SDAI at all visits
- 4. ACR20/50/70 response rates at all visits
- 5. Change from BL in individual components of ACR response at all visits
- Achievement of LDA at all visits. Low disease activity is defined as DAS28 (CRP) ≤ 3.2, DAS28(ESR) ≤ 3.2, CDAI ≤ 10, SDAI ≤ 11
- 7. Achievement of clinical remission at all visits. Clinical remission is defined as DAS28 (CRP) < 2.6, DAS28(ESR) < 2.6, CDAI ≤ 2.8, SDAI ≤ 3.3
- 8. Change in Short Form-36 (SF-36) from BL at Week 12
- Achievement of minimal clinically important difference (MCID) in change from BL in Health
   Assessment Questionnaire Disability Index (HAQ-DI) (defined as change from BL in Health
   Assessment Questionnaire ≤ -0.22) at all visits among subjects who have HAQ ≥ 0.22 at BL
- Achievement of response (such as LDA) based on DAS28 (CRP), CDAI, or SDAI over time from Week 12 to Week 24 among subjects who have achieved DAS28 (CRP), CDAI, or SDAI response at Week 12

Additional endpoint definitions are provided in Appendix D.

# 3.4 Safety Endpoints

The following safety evaluations will be performed during the study:



- 1. Treatment-emergent adverse events, serious adverse events (SAEs), adverse events (AEs) leading to discontinuation, AEs of special interest
- 2. Percent of subjects meeting potentially clinically significant criteria for vital signs, laboratory variables, physical examination findings and electrocardiogram (ECG) interval variables

# 3.5 Pharmacokinetic and Immunogenicity Endpoints

Serum or plasma concentrations of the conjugated ADC (ABBV-3373), total antibody, free payload A-1677770, and adalimumab (in the comparator arm) will be determined during the treatment period and drug washout period. If sufficient data are available from the optional intensive PK sampling group, terminal elimination half-life may be calculated and reported.

Anti-drug antibody (ADA) to either ABBV-3373 or adalimumab will be evaluated and if confirmed positive, titers will be measured. If required, samples will be analyzed for neutralizing antibodies (nAb).

# 3.6 Biomarker Endpoints

Biospecimens (e.g., blood, serum, and plasma) will be collected at specified time points (Appendix J) throughout the study to evaluate known and/or novel disease-related or drug-related biomarkers.

The analyses of biomarker samples will include but are not limited to proteins and genetic markers that will help to understand the subject's disease and response to study treatments. Changes in cortisol level under ABBV-3373 treatment and adalimumab will be assessed. Genes of interest will include those associated with PK, genes within the target pathway, or other genes believed to be related to RA and other inflammatory diseases. Samples for ribonucleic acid (RNA) and proteomics will be used to research if any genetic variants result in changes to gene expression or protein concentrations. Biomarker samples will be collected and analyzed from all subjects, unless precluded by local regulations or restrictions. For any samples collected in Germany, the research will be restricted to study drug and RA.

# 4 INVESTIGATIONAL PLAN

# 4.1 Overall Study Design and Plan

This is a randomized, double-blind, double-dummy, adalimumab active-controlled (12-week) Phase 2a study to assess the safety, tolerability, PK, pharmacodynamics, immunogenicity and efficacy following multiple IV administrations of ABBV-3373 or multiple SC injections of adalimumab in subjects with RA on background MTX. In the actively controlled period of the first 12 weeks of treatment, 45 subjects will receive either ABBV-3373 100 mg IV and the matching placebo for adalimumab SC eow or in the control arm the matching placebo for ABBV-3373 IV and adalimumab 80 mg SC eow (double-dummy) according to a 2:1 ratio. Thereafter all subjects enter a 12-week double-blind extension period. At Week 12, the administration of ABBV-3373 will stop (i.e., the last dose of ABBV-3373 will be given at Week 10) to assess the durability of the observed clinical effects up to 24 weeks. To keep blinding of the study beyond Week 12, the subjects randomized to ABBV-3373 will receive placebo injections, whereas



subjects randomized into the adalimumab arm will continue their 80 mg dosing until Week 22. At Week 12 and within the blinded extension period subjects who have not achieved at least a 20% improvement in both their swollen joint count (SJC) and tender joint count (TJC) based on 28 joint assessment compared with BL may be discontinued from the study at the discretion of the Investigator. Subsequently, standard of care may be administered at the discretion of the investigator.

After all endpoints are assessed at Week 24, a telephone contact is planned to follow up on safety 70 days after the last dose.

After all ongoing subjects complete the Week 12 study visit, the primary analysis for the ABBV-3373 cohort will be conducted to assess the primary/secondary endpoints and safety of this actively controlled period. A final analysis will be conducted after all subjects have completed Week 24 plus their safety follow-up. To maintain integrity of the trial, the study sites and subjects will remain blinded until the final analysis is completed.

The schematic of the study is shown in Figure 1. Further details regarding study procedures are located in Appendix K.



Figure 1. Study Schematic

 $\Delta DAS28(CRP)$  = change in disease activity score (DAS)28(C-reactive protein [CRP]); EOW = every other week; IV = intravenous; SC = subcutaneous



See Section 5.1 for information regarding eligibility criteria. See Section 5.8 for stratification factors for each cohort.

#### Pharmacokinetic Sampling

For ABBV-3373, blood samples for PK assessments will be collected according to the assessment schedule in Appendix J. Data from the first 12 subjects treated for at least 4 doses will be used in the PK interim analyses.

In addition, optional PK samples will be collected from subjects who consent to participate in the more intensive sampling group to provide data for PK characterization following repeated administrations. For these subjects, in addition to the standard sampling schedule, blood samples at the following time points will also be collected: Day 72, Day 73, Week 11, and Week 14.

# 4.2 Discussion of Study Design

#### **Choice of Control Group**

ABBV-3373 is an ADC, composed of adalimumab (the active component of Humira®) conjugated to A-1677770, a proprietary, highly potent GRM. In order to assess how the conjugation of adalimumab with the GRM impacts safety, tolerability and in particular whether it will provide additional efficacy versus (vs.) adalimumab, a direct comparison between the ADC and adalimumab is needed. The chosen study design with adalimumab as the positive control group allows such direct comparison. In addition, to compare clinical efficacy of the ADC with placebo control, and to address assay sensitivity, a synthetic placebo arm will be created with the propensity score matching approach using historical placebo subjects from similar trials with subject-level data.

#### Appropriateness of Measurements

Standard statistical, clinical, and laboratory procedures will be utilized in this study. All efficacy measurements in this study are standard for assessing disease activity in subjects with RA. All clinical and laboratory procedures in this study are standard and generally accepted.

#### Suitability of Subject Population

The specific population chosen was based on the unmet medical need of subjects as defined in Section 5.1.

#### Selection of Doses in the Study

Based on the clinical hypothesis, the ADC ABBV-3373 targets the activated immune cells that express transmembrane TNF to deliver the highly potent GRM selectively, therefore it has the potential to provide superior efficacy compared to a traditional anti-TNF antibody such as adalimumab. The dose of 100 mg IV eow for ABBV-3373 is selected to provide a similar systemic exposure to 80 mg adalimumab SC eow, which is a dose previously tested in RA subjects and twice as high as the recommended clinical regimen of 40 mg adalimumab SC eow. The rationale for selecting this higher dose is to increase tissue penetration of ABBV-3373 to successfully engage its intended target of transmembrane TNF on activated immune cells. Furthermore, the doses selected for ABBV-3373 and adalimumab are expected to generate similar systemic exposure to ensure a fair comparison between the two. Finally, 100 mg IV



ABBV-3373 is well within the range of doses that have been safely tested and well tolerated in the first-in-human SAD study. Historical data with adalimumab 80 mg eow or even higher in Phase 1 and 2 studies with adalimumab in the presence of  $MTX^{3,4}$  or 40 mg weekly as monotherapy in Phase 2 and 3 studies<sup>5,6</sup> have not shown any safety concerns.

#### **Study Duration**

For the patient population selected and the type of study drug tested, a 12-week primary endpoint to analyze the improvement of signs and symptoms and to assess the safety and tolerability of ABBV-3373 is appropriate. Preclinical data from a mouse collagen induced arthritis model<sup>2</sup> have shown a long lasting effect of the ADC in comparison to adequate control groups. Therefore, to assess the durability of the achieved clinical response at Week 12 in ABBV-3373-treated RA subjects, the subjects will be followed closely up to Week 24. While the maintenance of responses of ABBV-3373 will be monitored (under continuous placebo injections), subjects in the comparator arm will continue their adalimumab dosing to keep the blinding of the study.

#### 5 STUDY ACTIVITIES

# 5.1 Eligibility Criteria

Subjects must meet all of the following criteria in order to be included in the study. Anything other than a positive response to the questions below will result in exclusion from study participation.

#### Consent

1. Subjects or their legally authorized representative must voluntarily sign and date an informed consent, approved by an independent ethics committee (IEC)/institutional review board (IRB), prior to the initiation of any screening or study-specific procedures.

#### **Demographic and Laboratory Assessments**

- 2. Adult male or female, between 18 and 75 years of age inclusive at Screening.
- ② 3. Body mass index (BMI) is  $\ge 18.0$  to  $\le 39.9$  kg/m² after rounding to the nearest tenth. Body mass index is calculated as weight in kg divided by the square of height measured in meters.
- 4. Laboratory values meeting the following criteria within the screening period prior to the first dose of study drug:
  - Serum values of aspartate aminotransferase (AST) or alanine aminotransferase (ALT)
     < 2.5 × upper limit of normal (ULN);</li>
  - Absolute neutrophil count (ANC) > 1,500/μL;
  - Creatinine < 1.5 × ULN.</li>



- 5. Subject must have a negative test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg), HBc Ab (subjects who have been vaccinated against hepatitis B [HB] and are HBs Ab positive may be enrolled), hepatitis C virus (HCV) antibody (if Hepatitis C RNA level is undetectable at Screening, the subject can participate in this trial), and human immunodeficiency virus (HIV) Ab at Screening.
- 6. Subject is willing and able to comply with procedures required in this protocol.

#### **Diagnosis and Disease Activity**

- ▼ 7. Subject has the clinical diagnosis of RA for > 3 months based on the 1987 ACR classification criteria or 2010 ACR/European League against Rheumatism (EULAR) criteria.
- 8. Subject meets the following disease activity criteria: 
  ≥ 4 swollen joints (based on 28 joint count) and 
  ≥ 4 tender joints (based on 28 joint count) at Screening and BL Visits; and DAS28(CRP) 
  ≥ 3.2 at Screening.
- 9. Incomplete response to MTX. Subjects must have been on oral or parenteral MTX therapy
  ≥ 3 months and on a stable prescription of 15 to 25 mg/week (or ≥ 10 mg/week in subjects
  intolerant of MTX at doses ≥ 15 mg/week) for ≥ 4 weeks prior to the first dose of study drug.
  Subject must be expected to be able to continue on stable dose of MTX for the duration of study
  participation.

#### **Subject History**

- 10. Subject must not have been previously exposed to adalimumab or other anti-TNF biologics.
- 11. Subject <u>must not</u> have been previously exposed to non-anti-TNF biologics or targeted synthetic DMARDs for RA, with exception of subjects exposed for less than 3 months and terminated not due to lack of efficacy or intolerability.
- 12. No history of persistent chronic or active infection(s) requiring hospitalization or treatment with parenteral anti-infectives within 30 days, or oral anti-infectives within 14 days prior to the first dose of study drug administration.
- 13. No history of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
- 14. No history of moderate to severe congestive heart failure (CHF) (New York Heart Association Class III or IV).
- 15. No history or evidence of active TB disease or evidence of risk factors for latent TB infection OR a history of positive TB skin test or QuantiFERON-TB Gold In-Tube (GIT assay) within 90 days prior to study drug administration.
- 16. No history of pre-existing hyperglycemia (HbA1c > 6.5%), no history of osteoporotic fractures, and no high fracture risk (severe osteoporosis).
- 17. No history of pre-existing glaucoma, severe acne, osteonecrosis, uncontrolled hypertension, or peripheral edema.



- 18. No history of any malignancy except for successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix.
- 19. No history of clinically significant (per investigator's judgment) drug or alcohol abuse within
  the last 6 months.
- 20. <u>No history</u> of clinically significant medical conditions or any other reason that the investigator determines would **interfere with the subject's participation** in this study or would make the subject an unsuitable candidate to receive study drug.
- 21. No history of an allergic reaction or significant sensitivity to any constituents of the study drug, or an anaphylactic reaction to any agent (e.g., food products and bee sting), or a major reaction to any immunoglobulin G-containing product.
- 22. Is not currently enrolled in another clinical study, and has not been previously enrolled in this study.

#### Contraception

- 23. For all females of child-bearing potential; a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at BL prior to the first dose of study drug.
- 24. Female subjects of childbearing potential must practice at least 1 protocol-specified method of birth control, that is effective from Study Day 1 through at least 70 days after the last dose of study drug. Female subjects of non-childbearing potential do not need to use birth control.
- 25. Female who is not pregnant, breastfeeding, or considering becoming pregnant during the study or for approximately 70 days after the last dose of study drug.

#### **Concomitant Medications**

- 26. Subject must have discontinued all conventional synthetic disease-modifying antirheumatic drugs (csDMARDs), except for MTX. The washout periods for csDMARDs prior to the first dose of study are specified in Section 5.4.
- 27. Subject must not be on systemic GCs except for stable doses of GC (≤ 7.5 mg/d prednisone equivalent) in preceding 3 weeks prior to BL.
- 28. Subject <u>must not</u> have been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug.
- 29. Subject <u>must not</u> have been treated with any intra-articular, intramuscular, IV, trigger point or tender point, intra-bursa, or intra-tendon sheet corticosteroids in the preceding 8 weeks prior to the first dose of the study drug.
- 30. Subject <u>must not</u> have received any live vaccine within 4 weeks prior to the first dose of study drug, or expected need of live vaccination during study participation including at least 12 weeks after the last dose of study drug.



# 5.2 Contraception Recommendations

#### Contraception Requirements for Females

Subjects must follow the following contraceptive guidelines as specified:

#### Females, Non-Childbearing Potential

Females do not need to use birth control during or following study drug treatment if considered of non-childbearing potential due to meeting any of the following criteria:

- Postmenopausal, age > 55 years with no menses for 12 or more months without an alternative medical cause.
- Postmenopausal, age ≤ 55 years with no menses for 12 or more months without an alternative medical cause AND an FSH level > 40 IU/L.
- Permanently surgically sterile (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).

#### • Females, of Childbearing Potential

- Females of childbearing potential must avoid pregnancy while taking study drug(s) and for at least 70 days after the last dose of study drug.
- Females must commit to one of the following methods of birth control:
  - Combined (estrogen and progestogen containing) hormonal birth control (oral, intravaginal, transdermal, injectable) associated with inhibition of ovulation initiated at least 30 days prior to study BL Day 1.
  - Progestogen-only hormonal birth control (oral, injectable, implantable) associated with inhibition of ovulation initiated at least 30 days prior to study BL Day 1.
  - Bilateral tubal occlusion/ligation (can be via hysteroscopy, provided a hysterosalpingogram confirms success of the procedure).
  - Intrauterine device (IUD).
  - Intrauterine hormone-releasing system (IUS).
  - Vasectomized partner (provided the partner has received medical confirmation of the surgical success of the vasectomy and is the sole sexual partner of the trial subject).
  - Practice true abstinence, defined as: Refraining from heterosexual intercourse when
    this is in line with the preferred and usual lifestyle of the subject (periodic abstinence
    [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are
    not acceptable).

If required per local practices, male or female condom with or without spermicide OR cap, diaphragm or sponge with spermicide should be used in addition to one of the highly effective birth control methods listed above (excluding true abstinence).



Male subjects who are sexually active with a female partner of childbearing potential, must agree to use condoms, even if the male subject has undergone a successful vasectomy, from Study Day 1 through at least 70 days after the last dose of study drug.

Contraception recommendations related to use of concomitant therapies prescribed (e.g., MTX) should be based on the local label.

# 5.3 Prohibited Medications and Therapy

The following medications are prohibited throughout the duration of the study:

- Systemic GCs except stable doses of GC (≤ 7.5 mg/d prednisone equivalent) at BL, which have to be tapered off completely by end of Week 4.
- All csDMARDs, except MTX
- All targeted synthetic DMARDs: Examples include but are not limited to the following: Xeljanz® (tofacitinib), Olumiant® (baricitinib), Rinvoq® (upadacitinib)
- All biologic therapies. Examples include but are not limited to the following: Humira® (adalimumab), Enbrel® (etanercept), Remicade® (infliximab), Kineret® (anakinra), Rituxan® (rituximab), Cimzia® (certolizumab pegol), Simponi® (golimumab), Actemra® (tocilizumab), Raptiva® (efalizumab), Tysabri® (natalizumab), Stelara® (ustekinumab), Benlysta® (belimumab), Orencia® (abatacept), Prolia® (denosumab)
- Any intra-articular, intramuscular, parenteral, trigger point or tender point, intra-bursa, or intratendon sheet corticosteroids
- Any investigational drugs
- Any live vaccination

# 5.4 Prior and Concomitant Therapy

Any medication or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) that the subject is receiving at the time of enrollment or receives during the study must be recorded along with reasons for use; dates of administration, including start and end dates; and dosage information including dose, route, and frequency on the appropriate electronic case report form (eCRF) through the post-treatment contact (70 day follow-up call).

Non-Steroidal Anti-Inflammatory Drugs (NSAID) and low potency analgesics (i.e., tramadol, codeine, hydrocodeine, or propoxyphene) should continue to be used for the same reason and same dose each time but should not be taken within 24 hours prior to any study visit to avoid bias in outcome measurements.

Any questions regarding concomitant or prior therapy should be raised to the AbbVie emergency contact. Information regarding potential drug interactions with ABBV-3373 can be located in the ABBV-3373 Investigator's Brochure.<sup>2</sup>



Subjects must be able to safely discontinue any prohibited medications prior to initial study drug administration as specified in Section 5.1. Subjects must be consented for the study prior to discontinuing any prohibited medications for the purpose of meeting study eligibility.

Except for MTX, subject must have discontinued all csDMARDs. The washout period for csDMARDs prior to the first dose of study is specified below or should be at least five times the mean terminal elimination half-life of a drug.

- ≥ 4 weeks prior to first dose of study drug for minocycline, penicillamine, sulfasalazine, hydroxychloroquine, chloroquine, azathioprine, gold formulations, cyclophosphamide, tacrolimus, cyclosporine, mycophenolate or
- ≥ 8 weeks prior to first dose of study drug for leflunomide if no elimination procedure was followed, or adhere to an elimination procedure (i.e., 11 days with colestyramine, or washout with activated charcoal or as per local label).

If subjects have been exposed for less than 3 months with a non-anti-TNF biologic or targeted synthetic DMARD for RA and terminated not due lack of efficacy or intolerability, then it must be washed out for at least 5 half-lives.

#### Glucocorticoid Tapering of Subjects with ≤ 7.5 mg Prednisone Equivalent at BL

Up to 7.5 mg prednisone equivalent at BL is allowed. It is mandatory that subjects enrolling on concomitant GCs taper to discontinuation no later than completion of the Week 4 visit. Subjects may discontinue GCs prior to Week 4. If GC discontinuation during the first 4 weeks cannot be completed, the subject will be discontinued from the study; such subjects will be replaced.

The tapering scheme below can be considered a guide; adjustment may be required based on local availability of GC dose strengths (e.g., 5, 2.5, 2, 1 mg prednisone equivalents) and individual needs. If subjects enter with 6.5, 5.5, 4.5, 3.5, 2.5, or 1.5 mg/d then the tapering scheme for the next higher dose should be considered.

| Baseline (BL) | 7.5 or 7 mg/d | 6 mg/d | 5 mg/d | 4 mg/d | 3 mg/d | 2 mg/d |
|---------------|---------------|--------|--------|--------|--------|--------|
| BL to D7 | 5 | 4 | 2.5 | 2 | 2 | 1 |
| D8 to D14 | 5 | 4 | 2.5 | 2 | 2 | 1 |
| D15 to D21 | 2 | 2 | 1 | 1 | 1 | 1 |
| D22 to D29 | 2 | 2 | 1 | 1 | 1 | 1 |
| D30 onwards | 0 | 0 | 0 | 0 | 0 | 0 |

# 5.5 Withdrawal of Subjects and Discontinuation of Study

Subjects can request to be discontinued from participating in the study at any time for any reason including but not limited to disease progression or lack of response to treatment. The Investigator may discontinue any subject's participation at any time for any reason including but not limited to disease



progression, lack of response to treatment, an AE, safety concerns, or failure to comply with the protocol. See Section 6.2 for toxicity management criteria.

Subjects will have study drug discontinued immediately if any of the following occur:

- Clinically significant abnormal laboratory results or AEs, which rule out continuation of the study drug, as determined by the Investigator or the AbbVie Therapeutic Area Medical Director (TA MD).
- Serious infections (e.g., sepsis) that cannot be adequately controlled within 2 weeks by antiinfective treatment or would put the subject at risk for continued participation in the trial as determined by the Investigator.
- The Investigator believes it is in the best interest of the subject.
- The subject requests withdrawal from the study.
- Eligibility criteria violation was noted after the subject started study drug, when continuation of the study drug would place the subject at risk as determined by the AbbVie TA MD.
- Introduction of prohibited medications or dosages when continuation of the study drug would place the subject at risk, as determined by the AbbVie TA MD.
- Subject is non-compliant with TB prophylaxis (if applicable) or develops active TB at any time during the study.
- The subject becomes pregnant while on study drug.
- Malignancy, except for localized NMSC or carcinoma in-situ of the cervix.
- Subject is significantly non-compliant with study procedures which would put the subject at risk for continued participation in the trial as determined by the Investigator or the AbbVie TA MD.
- The subject develops anaphylactic reactions or anaphylactic shock.

In order to minimize missing data for efficacy and safety assessments, subjects who prematurely discontinue study participation should complete a Premature Discontinuation (PD) visit.

For subjects to be considered lost to follow-up, reasonable attempts must be made to obtain information on the subject's final status. At a minimum, 2 telephone calls must be made and 1 certified letter must be sent and documented in the subject's source documentation.

AbbVie may terminate this study prematurely, either in its entirety or at any site. The investigator may also stop the study at his/her site if he/she has safety concerns. If AbbVie terminates the study for safety reasons, AbbVie will promptly notify the investigator.

# 5.6 Follow-Up for Subject Withdrawal from Study

To minimize missing data for efficacy and safety assessments, subjects who prematurely discontinue study drug treatment should continue to be followed for all regularly scheduled visits, unless subjects have decided to discontinue the study participation entirely (withdrawal of informed consent). Subjects



should be advised on the continued scientific importance of their data even if they discontinue treatment with study drug early.

If a subject prematurely discontinues study participation (withdrawal of informed consent), the procedures outlined for the PD visit should be completed as soon as possible, preferably within 2 weeks. In addition, if subject is willing, a 70-day follow-up phone call after the last dose of study drug will be completed to ensure all treatment-emergent AEs/SAEs have been resolved.

All attempts must be made to determine the date of the last study drug dose and the primary reason for discontinuation of study drug or study participation. The information will be recorded on the appropriate eCRF page. However, these procedures should not interfere with the initiation of any new treatments or therapeutic modalities that the Investigator feels are necessary to treat the subject's condition. Following discontinuation of study drug, the subject should be treated in accordance with the Investigator's best clinical judgment irrespective of whether the subject decides to continue participation in the study.

#### Biomarker Research

In the event a subject withdraws consent from the clinical study, biomarker research will continue unless the subject explicitly requests analysis to be stopped. When AbbVie is informed that samples are withdrawn from research, samples will not be analyzed, no new biomarker analysis data will be collected for the withdrawn subject or added to the existing data or database(s). Data generated from clinical study and/or biomarker research, before subject withdrawal of consent, will remain part of the study results.

# 5.7 Study Drug

ABBV-3373 or matching placebo manufactured by AbbVie will be administered intravenously beginning on Day 1 (BL). Adalimumab or matching placebo manufactured by AbbVie will be administered subcutaneously beginning on Day 1 (BL). The administration of ABBV-3373 and matching placebo by venipuncture has to be given slowly over 15-30 minutes (via infusion line or infusion pump; the study drug can be diluted in 50-100 mL isotonic saline solution for this administration). Subjects have to be observed for at least 30 minutes thereafter.

AbbVie will provide study drug for ABBV-3373 or matching placebo and adalimumab or matching placebo. AbbVie-provided study drug should not be substituted or alternately sourced unless otherwise directed by AbbVie.

ABBV-3373 and matching placebo and adalimumab or matching placebo will be packaged in cartons with quantities sufficient to accommodate study design. Each kit will be labeled per local requirements and this label must remain affixed to the kit. Upon receipt, study drug should be stored as specified on the label and kept in a secure location. Each kit will contain a unique kit number. This kit number is assigned to a subject via interactive response technology (IRT) and encodes the appropriate study drug to be dispensed at the subject's corresponding study visit. Site staff will complete all blank spaces on the label before dispensing to subjects. Study drug will only be used for the conduct of this study.

AbbVie will provide instructions for drug preparation (Table 1).



Table 1. Identity of Investigational Product

| Study Drug | Dosage Form | Strength | Route of<br>Administration | Manufacturer |
|---|---|---|---|---|
| ABBV-3373 | Lyophilized powder<br>for solution for<br>infusion in vials | 50 mg/mL when reconstituted with 1.2 mL of sterile water for injection; 1 mL extractable volume per vial; further dilution into saline for IV infusion | IV | AbbVie |
| Placebo for ABBV-3373 | Lyophilized powder for solution for infusion in vials | N/A | IV | AbbVie |
| Adalimumab | Pre-filled syringe | 80 mg/0.8 mL | SC | AbbVie |
| Placebo for<br>Adalimumab | Pre-filled syringe | N/A | SC | AbbVie |

IV = intravenous; N/A = not applicable; SC = subcutaneous

# 5.8 Randomization/Drug Assignment

All subjects will be assigned a unique identification number by the IRT at the screening visit. For subjects who rescreen, the screening number assigned by the IRT at the initial screening visit should be used. The IRT will assign a randomization number that will encode the subject's treatment group assignment according to the randomization schedule generated by the statistics department at AbbVie.

Randomization will be stratified by factors listed in Section 4.1.

Forty-five subjects will be randomized to either the ABBV-3373 or adalimumab control arm according to a 2:1 ratio. Randomization will be stratified by the following factors:

- Stratification by current use of systemic GC (≤ 7.5 mg/d prednisone equivalent) for treatment of RA at BL (yes/no).
- Stratification by prior exposure to non-anti-TNF biologics or targeted synthetic DMARDs (< 3 months and terminated not due to lack of efficacy or intolerance) (yes/no).

All AbbVie personnel with direct oversight of the conduct and management of the trial (with the exception of AbbVie Drug Supply Management Team), the investigator, study site personnel, and the subject will remain blinded to each subject's treatment throughout the study. To maintain the blind, the ABBV-3373 vials and matching placebo vials, as well as adalimumab PFS and matching placebo PFS, will be provided for the study. The IRT will provide access to unblinded subject treatment information in the case of a medical emergency. The procedure for breaking the blind is referenced in the IRT Training Slides provided to each study site.



AbbVie must be notified before the blind is broken unless identification of the study drug is required for medical emergency, i.e., situation in which the knowledge of the specific blinded treatment will affect the immediate management of the subject/patient's conditions (e.g., antidote is available). AbbVie must then be notified within 24 hours of the blind being broken. See Appendix K for contact information, including 24/7 AbbVie emergency contact coverage.

#### 5.9 Protocol Deviations

The investigator is responsible for complying with all protocol requirements, written instructions, and applicable laws regarding protocol deviations. Protocol deviations are prohibited except when necessary to eliminate an immediate hazard to study subjects. If a protocol deviation occurs (or is identified), the investigator is responsible for notifying IEC/independent review board (IRB), regulatory authorities (as applicable), and AbbVie.

#### 6 SAFETY CONSIDERATIONS

### 6.1 Complaints and Adverse Events

#### Complaints

A complaint is any written, electronic, or oral communication that alleges deficiencies related to the physical characteristics, identity, quality, purity, potency, durability, reliability, safety, effectiveness, or performance of a product/device. Complaints associated with any component of this investigational product must be reported to AbbVie.

#### **Product Complaint**

A product complaint is any complaint related to the biologic or drug component of the product or to the medical device component(s).

For a product this may include, but is not limited to, damaged/broken product or packaging, product appearance whose color/markings do not match the labeling, labeling discrepancies/inadequacies in the labeling/instructions (e.g., printing illegible), missing components/product, device not working properly, or packaging issues.

Product complaints concerning the investigational product and/or device must be reported to AbbVie within 1 business day of the study site's knowledge of the event. Product complaints occurring during the study will be followed up to a satisfactory conclusion.

#### Medical Complaints/Adverse Events and Serious Adverse Events

An AE is defined as any untoward medical occurrence in a subject or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.



The investigators will monitor each subject for clinical and laboratory evidence of AEs on a routine basis throughout the study. All AEs will be followed to a satisfactory conclusion.

An elective surgery/procedure scheduled to occur during a study will not be considered an AE if the surgery/procedure is being performed for a pre-existing condition and the surgery/procedure has been pre planned prior to study entry. However, if the pre-existing condition deteriorates unexpectedly during the study (e.g., surgery performed earlier than planned), then the deterioration of the condition for which the elective surgery/procedure is being done will be considered an AE.

If any of the following SAEs or AEs are reported, then the following supplemental report must be completed.

| Serious Adverse Event | Supplemental Report |
|---|---|
| Cardiac events Myocardial infarction or unstable angina Heart failure Cerebral vascular accident and transient ischemic attack Cardiovascular procedures (SAE Supplemental Procedure eCRF) | MACE eCRF |
| Discontinuation or interruption of study drug due to a hepatic-related AE A hepatic-related SAE ALT/AST > 8 × ULN or ALT/AST > 3 × ULN with a total bilirubin > 2 × ULN | Hepatic AE eCRF |

AE = adverse event; ALT = alanine aminotransferase; AST = aspartate aminotransferase; eCRF = electronic Case Report Form; MACE = major adverse cardiac event; SAE = serious adverse event; ULN = upper limit of normal

If an AE, whether associated with study drug or not, meets any of the following criteria, it is to be reported to AbbVie clinical pharmacovigilance or contract research organization (as appropriate) as a SAE within 24 hours of the site being made aware of the SAE (refer to Section 4.3 of the Operations Manual for reporting details and contact information):

| Death of Subject | An event that results in the death of a subject. |
|---|---|
| Life-Threatening | An event that, in the opinion of the investigator, would have resulted in immediate fatality if medical intervention had not been taken. This does not include an event that would have been fatal if it had occurred in a more severe form. |
| Hospitalization or<br>Prolongation of<br>Hospitalization | An event that results in an admission to the hospital for any length of time or prolongs the subject's hospital stay. This does not include an emergency room visit or admission to an outpatient facility. |
| Congenital Anomaly | An anomaly detected at or after birth, or any anomaly that results in fetal loss. |



# Persistent or Significant Disability/Incapacity

An event that results in a condition that substantially interferes with the activities of daily living of a study subject. Disability is not intended to include experiences of relatively minor medical significance such as headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle).

Important Medical Event Requiring Medical or Surgical Intervention to Prevent Serious Outcome An important medical event that may not be immediately life-threatening or result in death or hospitalization, but based on medical judgment may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above (i.e., death of subject, life threatening, hospitalization, prolongation of hospitalization, congenital anomaly, or persistent or significant disability/incapacity). Additionally, any elective or spontaneous abortion or stillbirth is considered an important medical event. Examples of such events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

All adverse events reported from the time of study drug administration until 70 days after discontinuation of study drug administration will be collected, whether solicited or spontaneously reported by the subject. In addition, serious adverse events and protocol-related nonserious adverse events will be collected from the time the subject signs the study-specific informed consent.

AbbVie will be responsible for Suspected Unexpected Serious Adverse Reactions (SUSAR) reporting for the Investigational Medicinal Product (IMP) in accordance with global and local requirements.

Adverse events will be monitored throughout the study to identify any of special interest that may indicate a trend or risk to subjects.

#### Serious Adverse Event Reporting

AbbVie is committed to continue to collect safety information including those events that may occur in this trial in order to confirm this established safety profile and to identify any unknown potential adverse reactions, rare events, and those events with a long latency. AbbVie is participating in a Food and Drug Administration-requested, TNF inhibitor class wide exploration of the rare appearance of malignancy in subjects/patients who are 30 years of age or younger at the time of diagnosis. The risk of malignancy in this age group has not been established and is difficult to study due to its rarity. AbbVie appreciates your attention to the additional reporting requirements needed in this unlikely event. In the event of an SAE, and additionally, any nonserious event of malignancy in subjects 30 years of age and younger, whether related to SC study drug or not, the physician will notify Clinical Pharmacovigilance within 24 hours of the physician becoming aware of the event by entering the SAE or nonserious event of malignancy in subjects 30 years of age and younger data into the electronic data capture (EDC) system. Serious adverse events and nonserious events of malignancy in subjects 30 years of age and younger, that occur prior to the site having access to the RAVE® EDC system or if RAVE® is not operable, should be documented on the SAE non-case report form forms and emailed (preferred route) or faxed to the Clinical Pharmacovigilance within 24 hours of being made aware of the SAE.



#### Adverse Events of Special Interest

The following adverse events of special interest will be monitored during the study:

- Serious infections, opportunistic infections, herpes zoster, and TB;
- Malignancy (all types);
- Cardiovascular events (e.g., major adverse cardiovascular event [MACE]);
- Hematologic disorders (i.e., anemia, neutropenia, lymphopenia);
- Hepatic disorders;
- Hypersensitivity reactions, including all serious allergic reactions;
- Demyelinating disease;
- Systemic GC side effects (i.e., infections, skin atrophy, weight gain, cataract, hypertension, indigestion, hyperglycemia).

#### Adverse Event Severity and Relationship to Study Drug

The investigator will classify AEs according to the Rheumatology Common Toxicity Criteria v.2.0 (Appendix I).

The investigator will use the following definitions to assess the relationship of the AE to the use of study drug:

**Reasonable Possibility** After consideration of factors including timing of the event, biologic

plausibility, clinical judgment, and potential alternative causes, there is sufficient evidence (information) to suggest a causal relationship.

sufficient evidence (information) to suggest a causal relationship.

**No Reasonable Possibility** After consideration of factors including timing of the event, biologic

plausibility, clinical judgment, and potential alternative causes, there is insufficient evidence (information) to suggest a causal relationship.

#### Pregnancy

While not an AE, pregnancy in a study subject must be reported to AbbVie within 1 working day after the site becomes aware of the pregnancy. Subjects who become pregnant during the study must be discontinued (Section 5.5). If a pregnancy occurs in a study subject or in the partner of a study subject, information regarding the pregnancy and the outcome will be collected.

In the event of pregnancy occurring in a subject's partner during the study, written informed consent from the partner must be obtained prior to collection of any such information. AbbVie will provide a separate consent form for this purpose. Pregnancy in a subject's partners will be collected from the date of the first dose through 70 days following the last dose of study drug.

The pregnancy outcome of an elective or spontaneous abortion, stillbirth or congenital anomaly is considered a SAE and must be reported to AbbVie within 24 hours after the site becomes aware of the event.



# 6.2 Toxicity Management

The management of specific AEs and laboratory parameters is described in Table 2 and in the Operations Manual (Appendix K).

The toxicity management of the AEs including AEs of special interest consists of safety monitoring (review of AEs on an ongoing basis, and periodical/ad hoc review of safety issues by a safety data monitoring committee), interruption of study drug dosing with appropriate clinical management if applicable, and discontinuation of the subjects from the study drug. The management of specific AEs and laboratory parameters is described below.

For subjects who discontinued study drug but continued study participation and are on standard of care therapies, these toxicity management requirements do not apply (including alerts from the central lab) and any intolerability to standard of care therapies should be managed by the prescribing physician.

#### Management of Hypersensitivity and Serious Allergic Reactions

Subjects should be closely monitored and assessed for the development of signs and symptoms of hypersensitivity reactions, including anaphylaxis. Drug administration (ABBV-3373) should be done slowly over 15 - 30 minutes (via infusion line or infusion pump; the study drug can be diluted in 50 - 100 mL isotonic saline solution for this administration), and subjects should be observed for at least 30 minutes thereafter. Study drug should be discontinued and appropriate therapy be instituted if a subject develops clinically significant hypersensitivity reactions.

#### Hypersensitivity Testing

In the event of a suspected systemic post-dose hypersensitivity reaction, if the clinical situation allows, every effort should be made to obtain a serum sample within 2 hours but no later than 6 hours from symptom onset for additional blood tests (e.g, tryptase, ADA, nAb, total IgE, total hemolytic complement, etc.). Additional details regarding hypersensitivity testing can be found in the Operations Manual, Section 3.12 (Appendix K).

#### Management of Serious Infections

Subjects should be closely monitored for the development of signs and symptoms of infection during and after treatment with study drug. Study drug should be interrupted if a subject develops a serious infection or a serious opportunistic infection. A subject who develops a new infection during treatment with study drug should undergo prompt diagnostic testing appropriate for an immunocompromised subject. As appropriate, antimicrobial therapy should be initiated, and the subject should be closely monitored. Study drug may be restarted once the infection has been successfully treated. Subjects who develop active TB must be permanently discontinued from study drug.

#### Management of Malignancy

Subjects who develop malignancy other than NMSC or carcinoma in-situ of the cervix must be discontinued from the study drug. Information including histopathological results should be queried for the confirmation of the diagnosis.



#### Management of Demyelinating Disease

Subjects must be discontinued from study drug with new onset or exacerbation of clinical symptoms and/or radiographic evidence of central nervous system demyelinating disease (including multiple sclerosis), optic neuritis, and peripheral demyelinating disease (including Guillain Barré syndrome).

#### Management of Hypertension

Subjects should be closely monitored for the development of hypertension before and 30 minutes after treatment with study drug. Study drug should be interrupted if a subject develops serious hypertension in which case they should be monitored under standard of care.

#### Management of Hyperglycemia

Subjects should be closely monitored for the development of hyperglycemia during and after treatment with study drug. Study drug should be interrupted if a subject develops a serious hyperglycemia in which case they should be monitored under standard of care.

#### Management of GC-Induced Adrenal Insufficiency

High dose or long term use of corticosteroids can produce reversible HPA axis suppression with the potential for GC insufficiency after withdrawal of treatment. Drug-induced secondary adrenocortical insufficiency may be minimized by gradual reduction of dosage. This type of relative insufficiency may persist for months after discontinuation of therapy; therefore, hormone therapy should be reinstituted in any situation of stress occurring during that period.

#### Management of Select Laboratory Abnormalities

For any given laboratory abnormality, the investigator should assess the subject, apply the standard of care for medical evaluation and treatment following any local guidelines. Specific toxicity management guidelines for selected abnormal laboratory values are described in Table 2, and may require a supplemental eCRF to be completed (Section 6.1 [Complaints and AEs]). All abnormal laboratory tests that are considered clinically significant by the investigator will be followed to a satisfactory resolution. If a repeat test is required per Table 2, the repeat testing must occur as soon as possible.

Table 2. Specific Toxicity Management Guidelines for Abnormal Laboratory Values

| Laboratory<br>Parameter | Toxicity Management Guideline |
|---|---|
| Hemoglobin | If hemoglobin < 8 g/dL interrupt study drug dosing and confirm by repeat testing with new sample |
| | <ul> <li>If hemoglobin decreases ≥ 3.0 g/dL from BL, without an alternative etiology,<br/>interrupt study drug dosing and confirm by repeat testing with new sample.</li> </ul> |
| | • If hemoglobin decreases ≥ 3.0 g/dL from BL and an alternative etiology is known, the subject may remain on study drug at the investigator's discretion. |
| | If confirmed, continue to withhold study drug until hemoglobin value returns to normal reference range or its BL value. |



| Laboratory<br>Parameter | Toxicity Management Guideline |
|---|---|
| Absolute neutrophil count (ANC) | <ul> <li>If confirmed &lt; 1000/μL by repeat testing with new sample, interrupt study drug<br/>dosing until ANC value returns to normal reference range or its BL value.</li> </ul> |
| | • Discontinue study drug if confirmed < 500/μL by repeat testing with new sample. |
| Absolute<br>lymphocyte counts<br>(ALC) | <ul> <li>If confirmed &lt; 500/μL by repeat testing with new sample, interrupt study drug<br/>dosing until ALC returns to normal reference range or its BL value.</li> </ul> |
| Total white blood cell count | <ul> <li>If confirmed &lt; 2000/μL by repeat testing with new sample, interrupt study drug<br/>dosing until white blood cell count returns to normal reference range or its BL value.</li> </ul> |
| Platelet count | <ul> <li>If confirmed &lt; 50,000/μL by repeat testing with new sample, interrupt study drug<br/>dosing until platelet count returns to normal reference range or its BL value.</li> </ul> |
| AST or ALT | <ul> <li>Interrupt study drug if confirmed ALT or AST &gt; 3 × ULN by repeat testing with new sample and either a total bilirubin &gt; 2 × ULN or an international normalized ratio (INR) &gt; 1.5.</li> </ul> |
| | <ul> <li>A separate blood sample for INR testing will be needed to measure INR at the<br/>time of repeat testing for ALT or AST. A repeat test of INR is not needed for<br/>determination if above toxicity management criteria are met.</li> </ul> |
| | • Interrupt study drug if confirmed ALT or AST > 3 × ULN by repeat testing with new sample along with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%). |
| | <ul> <li>Interrupt study drug if confirmed ALT or AST &gt; 5 × ULN by repeat testing with new<br/>sample for more than 2 weeks.</li> </ul> |
| | <ul> <li>Interrupt study drug if confirmed ALT or AST &gt; 8 × ULN by repeat testing with new<br/>sample.</li> </ul> |
| | Subjects who meet any of the above criteria should be evaluated for an alternative etiology of the ALT or AST elevation and managed as medically appropriate. The investigator should contact the AbbVie TA MD to discuss the management of a subject when an alternative etiology has been determined. The alternative etiology should be documented appropriately in the eCRF; study drug should be discontinued if no alternative etiology can be found and ALT or AST elevations persist. |
| | For any confirmed ALT or AST elevations > 3 ULN, complete the appropriate supplemental hepatic eCRF(s). |
| | Subjects with HBc Ab+ (irrespective of HBs Ab status) and negative HBV DNA PCR testing at Screening who develop the following should have HBV DNA PCR testing performed within one week: |
| | • ALT > 5 × ULN OR |
| | ALT or AST > 3 × ULN and either a total bilirubin > 2 × ULN or INR > 1.5 OR |
| | ALT or AST > 3 × ULN along with clinical signs of possible hepatitis. A positive result for UDV DNA DCD testing will require interest distaint which is to require in the positive result for UDV DNA DCD testing will require interest distaint which is to require in the positive requirement. |
| | A positive result for HBV DNA PCR testing will require immediate interruption of study drug (unless not acceptable by local practices) and a hepatologist consultation should occur within 1 week for recommendation regarding subsequent treatment. |



| Laboratory<br>Parameter | Toxicity Management Guideline |
|---|---|
| Serum Creatinine | <ul> <li>If serum creatinine is &gt; 1.5 × the BL value and &gt; ULN, repeat the test for serum creatinine (with subject in an euvolemic state) to confirm the results. If the results of the repeat testing still meet this criterion, then interrupt study drug and re-start study drug once serum creatinine returns to ≤ 1.5 × BL value and ≤ ULN.</li> <li>For the above serum creatinine elevation scenario, complete the appropriate supplemental renal eCRF(s).</li> </ul> |
| Creatine<br>Phosphokinase<br>(CPK) | <ul> <li>If confirmed CPK value ≥ 4 × ULN and there are no symptoms suggestive of myositis<br/>or rhabdomyolysis, the subjects may continue study drug at the investigator's<br/>discretion.</li> </ul> |
| | <ul> <li>If CPK ≥ 4 × ULN accompanied by symptoms suggestive of myositis or<br/>rhabdomyolysis, interrupt study drug and contact AbbVie TA MD.</li> </ul> |
| | For the above CPK elevation scenarios, complete supplemental increased CPK eCRF. |

Ab = antibody; ALC = Absolute lymphocyte counts; ALT = alanine aminotransferase; ANC = absolute neutrophil count; AST = aspartate aminotransferase; BL = baseline; CPK = creatine phosphokinase; DNA = deoxyribonucleic acid; eCRF = electronic case report form; HB = hepatitis B; HBV = hepatitis B virus; INR = international normalized ratio; PCR = polymerase chain reaction; TA MD = Therapeutic Area Medical Director; ULN = upper limit of normal

#### Management of ECG Abnormality

Subjects should be discontinued for an ECG change considered clinically significant OR a confirmed absolute QT interval corrected for heart rate using Fridericia's correction formula (QTcF) value > 500 msec.

# 7 STATISTICAL METHODS & DETERMINATION OF SAMPLE SIZE

# 7.1 Statistical and Analytical Plans

The statistical methods provided in this protocol will be focused on primary and secondary analyses. Complete and specific details of the statistical analysis will be described in the Statistical Analysis Plan (SAP). All statistical analyses will be performed using SAS (SAS Institute Inc., Cary, North Carolina, USA).

# 7.2 Definition for Analysis Populations

The Full Analysis Set (FAS) includes all randomized subjects who received at least 1 dose of the study drugs. The FAS will be used for all efficacy analyses. Subjects will be grouped according to treatment as randomized. The Per-Protocol Analysis Set represents a subset of the FAS and consists of all FAS subjects without any major violations. Additional analysis may be conducted on the Per-Protocol Analysis Set as deemed appropriate, in order to evaluate the impact of major protocol violations on the primary endpoint.



The Safety Analysis Set consists of all subjects who received at least 1 dose of the study drugs. For the Safety Analysis Set, subjects are grouped based on the treatment actually received, regardless of the treatment randomized.

# 7.3 Statistical Analyses for Efficacy

#### **Primary Endpoint Analysis**

Analysis of the primary endpoint will be conducted on the FAS based on treatment as randomized.

The primary endpoint is the change from BL in DAS28(CRP) at Week 12. The historical mean and standard deviation of the change from BL in DAS28(CRP) at Week 12 in adalimumab 80 mg eow are estimated to be –2.13 and 1.35 respectively based on a meta-analysis of 3 historical adalimumab studies (Studies DE007, DE009, and DE011).

The first comparison in order to achieve the first primary objective of assessing the efficacy of ABBV-3373 is to compare change from BL in DAS28(CRP) at Week 12 in the ABBV-3373 group with –2.13, the adalimumab 80 mg eow historical mean change from BL at Week 12 based on the meta-analysis. The treatment mean change from BL and 90% confidence interval of ABBV-3373 will be estimated from Mixed Effect Model Repeated Measurements (MMRM) method including up to Week 12 data with treatment group, visits, treatment-by-visit interaction, BL values of the primary endpoint, and stratification factors with observed case (OC) data. The study will be declared positive if the comparison is significant and favoring ABBV-3373.

In order to achieve the second primary objective of comparing clinical efficacy of ABBV-3373 with adalimumab and to test the concept that an anti-TNF ADC has the potential to provide superior efficacy than the traditional anti-TNF antibody in RA, the second comparison is to compare ABBV-3373 with adalimumab for the primary efficacy endpoint with a Bayesian historical data borrowing approach. The same MMRM model as described in the first comparison will be used to estimate in-study mean and standard deviation. Informative normal prior for adalimumab will be determined based on historical adalimumab data and a non-informative prior will be used for ABBV-3373. The prior distributions and estimates from MMRM model will be combined to construct the posterior distributions which will be used for comparison between ABBV-3373 and adalimumab.

If the adalimumab group mean is not comparable with historical adalimumab data, for example, the confidence intervals of the mean based on historical and in-trial data don't overlap, the Bayesian approach based on historical data will not be performed, and the mean difference in change from BL in DAS28(CRP) at Week 12 between the ABBV-3373 group and adalimumab will be estimated only based on in-study data with the MMRM model described above.

Historical data borrowing will only apply to the primary endpoint.

To address the secondary objectives of assay sensitivity, a synthetic placebo arm will be created with the propensity score matching approach using historical placebo subjects from similar trials with subject-level data. Details will be provided in the SAP.



#### Secondary Endpoints and Additional Endpoints Analyses for BL to Week 12

For the first 12 weeks of treatment period, continuous efficacy variables will be analyzed using an MMRM method. Categorical efficacy variables will be analyzed using the Cochran-Mantel-Haenszel (CMH) test controlling for stratification variables. Non-responder imputation (NRI) will be used for primary inference purpose. Observed Case data will be summarized descriptively as a sensitivity analysis.

#### Additional Endpoints Analyses up to Week 24

Statistical inference of additional continuous endpoints at each visit up to Week 24 will be conducted using analysis of covariance (ANCOVA) with treatment and stratification factors as the fixed factors and the corresponding BL value as the covariate. Additional categorical efficacy variables up to Week 24 will be analyzed using the same CMH test as for the binary secondary endpoint analysis.

Details on the analyses of the primary and other efficacy endpoints will be provided in the SAP.

#### Sample Size Estimation

The primary endpoint is the mean change of DAS28(CRP) from BL at Week 12. Two comparisons are considered. The first one is to compare mean change in DAS28(CRP) of the ABBV-3373 group to that of historical adalimumab 80 mg eow, which is -2.13. Assuming a mean DAS28(CRP) change from BL of -2.769 to -2.982 for ABBV-3373 (corresponding to 30% to 40% more reduction than historical adalimumab) and a standard deviation of 1.35, 30 subjects on ABBV-3373 will provide an approximate 81% to 96% power with a one-sample t-test and one-sided alpha = 0.05 significance level.

The second comparison is between ABBV-3373 arm and adalimumab arm with borrowed historical adalimumab data using a Bayesian approach. When considering borrowing historical data, the planned sample size is 45 subjects (30 in ABBV-3373 and 15 in adalimumab). The study will be considered successful if the posterior probability of mean difference < 0 is larger than 95%, i.e.,:

$$P(\mu_{ABBV-3373} - \mu_{Adalimumab} < 0|data) > 0.95.$$

Based on the historical mean and standard deviation from adalimumab meta-analysis, a prior distribution for adalimumab is N (-2.13,  $0.246^2$ ) corresponding to the 30 historical subjects borrowed. A noninformative prior for ABBV-3373 treatment group will be set. Given the mean change from BL in DAS28 (CRP) is -2.13 for adalimumab, the probability to claim the study success is approximately 66% to 88% if the mean change from BL in DAS28 (CRP) is -2.769 to -2.982 for ABBV-3373 (i.e., 30% to 40% more reduction than historical adalimumab), with at least 45 subjects for adalimumab (15 in-trial and at least 30 borrowed) and 30 subjects for ABBV-3373. If both ABBV-3373 and adalimumab groups have the same mean change from BL of -2.13, the probability to claim study success (equivalent to type I error rate) is approximately 0.03 with the same sample sizes. In the event that adalimumab variability precludes historic data borrowing, using only the in-study 15 adalimumab subjects and 30 ABBV-3373 subjects will provide 43% to 63% power when ABBV-3373 in 30% to 40% more reduction than adalimumab respectively.



# 7.4 Statistical Analyses for Safety

Safety analyses will be carried out using the Safety Analysis Set. There will be 2 sets of planned safety analyses: safety analysis by Week 12 and long-term safety analysis. Safety will be assessed by AEs, laboratory assessments, and vital signs. Frequency tables of subjects with treatment emergent AEs by preferred term (PT), by system organ class (SOC) and PT as in the Medical Dictionary for Regulatory Activities, by severity, and by relationship to the study drug as assessed by the Investigator will be provided.

Summaries of SAEs, deaths, AEs leading to discontinuation, and Areas of Safety Interest will be provided as well. The changes from BL in clinical laboratory and vital sign values by visit will be analyzed in a descriptive manner. Shift of selected laboratory values from BL to defined time points will be tabulated. The number and percentage of subjects meeting the criteria for potentially clinically significant laboratory/vital sign/ physical examination/ECG values will be summarized.

No external data borrowing will be applied for safety analyses.

# 7.5 Statistical Analysis of Pharmacokinetic and Immunogeniticy Data

Concentrations of conjugated ADC (ABBV-3373), total antibody, free payload A-1677770, and adalimumab (in the comparator arm), along with all applicable PK parameters will be summarized at each time point for each group using descriptive statistics.

Population PK analyses combining the data from this study and other studies may be performed and reported outside of the clinical study report.

Anti-drug antibody and nAb incidence and ADA titer values will be summarized for each group using descriptive statistics.

# 7.6 Statistical Analysis of Biomarker Data

Analysis will be conducted on biomarker data for the purpose of identification of prognostic, predictive, surrogate, and pharmacodynamic biomarkers associated with efficacy or safety. The association of biomarkers to the efficacy or safety endpoints will be explored for each biomarker one at a time, and also for combinations of biomarkers via some multivariate predictive modeling approaches.

# 7.7 Interim Analysis

An interim PK analysis after 12 subjects are treated for at least 4 doses will be performed to assess whether the observed total antibody systemic exposure following ABBV-3373 administration is in the approximate range of 80 mg adalimumab exposure based on trough concentration ( $C_{trough}$ ) levels and if there is a need for dose adjustment for ABBV-3373 and replacement of already-treated subjects.



#### 8 ETHICS

# 8.1 Independent Ethics Committee/Institutional Review Board (IEC/IRB)

The protocol, informed consent form(s), recruitment materials, and all subject materials will be submitted to the IEC/IRB for review and approval. Approval of both the protocol and the informed consent form(s) must be obtained before any subject is enrolled. Any amendment to the protocol will require review and approval by the IEC/IRB before the changes are implemented to the study. In addition, all changes to the consent form(s) will be IEC/IRB approved.

# 8.2 Ethical Conduct of the Study

The study will be conducted in accordance with the protocol, Operations Manual, International Council for Harmonisation (ICH) guidelines, applicable regulations, and guidelines governing clinical study conduct and the ethical principles that have their origin in the Declaration of Helsinki. Responsibilities of the investigator are specified in Appendix B.

# 8.3 Subject Confidentiality

To protect subjects' confidentiality, all subjects and their associated samples will be assigned numerical study identifiers or "codes." No identifiable information will be provided to AbbVie.

# 9 SOURCE DOCUMENTS AND CASE REPORT FORM COMPLETION

The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. All source documents should be attributable, legible, contemporaneous, original, accurate, and complete to ensure accurate interpretation of data. Clinical site monitoring is conducted to ensure that the rights and well-being of human subjects are protected, that the reported trial data are accurate, complete, and verifiable, and that the conduct of the trial is in compliance with the currently approved protocol, ICH Good Clinical Practice (GCP), and applicable local regulatory requirement(s).

# 10 DATA QUALITY ASSURANCE

AbbVie will ensure that the clinical trial is conducted with a quality management system that will define quality tolerance limits in order to ensure human subject protection and reliability of study results. Data will be generated, documented, and reported in compliance with the protocol, ICH GCP, and applicable regulatory requirements.



# 11 COMPLETION OF THE STUDY

The end-of-study is defined as last subject last visit (70 day follow-up call).

#### 12 REFERENCES

- 1. Schäcke H, Döcke WD, Asadullah K. Mechanisms involved in the side effects of glucocorticoids. Pharmacol Ther. 2002;96(1):23-43.
- 2. AbbVie. ABBV-3373 Investigator's Brochure Edition 3. September 2019. Addendum 1, Edition 3. November 2019.
- 3. Keystone E, Weinblatt M, Furst D, et al. Adalimumab, a fully human anti-TNF monoclonal antibody  $\alpha$  monoclonal antibody, for treatment of rheumatoid arthritis in patients taking concomitant methotrexate: The ARMADA trial. Arthritis Rheum. 2003;48(1):35-45.
- 4. Weisman M, Keystone E, Paulus H, et al. A dose escalation study designed to demonstrate the safety, tolerability and efficacy of the fully human anti-TNF antibody, D2E7, given in combination with methotrexate (MTX) in patients with active RA (abstract 1948). Arthritis Rheum. 2000;43(9):S391.
- 5. van de Putte LBA, Rau R, Breedveld F, et al. Efficacy and safety of the fully human anti-tumour necrosis factor  $\alpha$  monoclonal antibody adalimumab (D2E7) in DMARD refractory patients with rheumatoid arthritis: a 12 week, phase II study. Ann Rheum Dis. 2003;62(12):1168-77.
- 6. van de Putte LB, Atkins C, Malaise M, et al. Efficacy and safety of adalimumab as monotherapy in patients with rheumatoid arthritis for whom previous disease modifying anti-rheumatic drug treatment has failed. Ann Rheum Dis. 2004;63(5):508-16.



# APPENDIX A. STUDY SPECIFIC ABBREVIATIONS AND TERMS

| Abbreviation | Definition |
|--------------|------------|
|--------------|------------|

ACR American College of Rheumatology

ACR20 American College of Rheumatology 20% improvement criteria
ACR50 American College of Rheumatology 50% improvement criteria

ADA anti-drug antibody

ADC antibody-drug conjugate
ADL activities of daily living

AE adverse event

ALT alanine aminotransferase

ANC absolute neutrophil count

ANCOVA analysis of covariance

AST aspartate aminotransferase

BL baseline

BMI body mass index

CDAI clinical disease activity index
CHF congestive heart failure

CMH Cochran-Mantel-Haenszel

CR clinical remission
CRF case report form
CRP C-reactive protein

csDMARD conventional synthetic disease-modifying antirheumatic drug

Ctrough trough concentration measured at the end of a dosing interval at steady state

DAS disease activity score

DAS28 disease activity score (28 joints)

DMARD disease-modifying antirheumatic drug

DNA deoxyribonucleic acid
ECG electrocardiogram

eCRF electronic case report form
EDC electronic data capture

eow every other week

ESR erythrocyte sedimentation rate

EULAR European League Against Rheumatism


FAS full analysis set

FSH follicle-stimulating hormone

GC glucocorticoid

GCP good clinical practice

GRMs glucocorticoid receptor modulators

HAQ-DI Health Assessment Questionnaire Disability Index

HAV hepatitis A virus

HAV-IgM hepatitis A virus immunoglobulin M

HB hepatitis B

HBsAg hepatitis B surface antigen

HBV hepatitis B virus
HCV hepatitis C virus

HIV human immunodeficiency virus
HPA hypothalamic-pituitary-adrenal

hs-CRP high-sensitivity C-reactive protein

ICH International Council for Harmonisation

IEC Independent ethics committee

IL interleukin

IMP Investigational Medicinal Product

IRB institutional review board

IRT interactive response technology

IUD intrauterine device

IUS intrauterine hormone-releasing system

IV intravenous

LDA low disease activity

MACE major adverse cardiac event

MCID minimal clinically important difference

MedDRA Medical Dictionary for Regulatory Activities

MMRM Mixed Effect Model Repeated Measurements

MTX Methotrexate

nAb neutralizing antibody

NMSC non-melanoma skin cancer

NRI non-responder imputation

NSAID nonsteroidal anti-inflammatory drug



OC observed case

QT interval corrected for heart rate using Fridericia's correction formula

PD premature discontinuation

PK pharmacokinetic(s)
PT preferred term

RA rheumatoid arthritis

RNA ribonucleic acid

SAD single ascending dose
SAE serious adverse event
SAP statistical analysis plan

SC subcutaneous

SDAI simplified disease activity index
SF-36 36-Item Short Form Health Survey

SJC swollen joint count
SOC system organ class

SUSAR suspected unexpected serious adverse reactions

TA MD Therapeutic Area Medical Director

TB tuberculosis

TJC tender joint count

TNF tumor necrosis factor
ULN upper limit of normal
VAS visual analogue scale

vs. versus



## APPENDIX B. RESPONSIBILITIES OF THE INVESTIGATOR

Protocol M16-560: A Randomized, Double-Blind, Double-Dummy, Active Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABBV-3373 in Subjects with Moderate to Severe Rheumatoid Arthritis

Protocol Date: 04 September 2020

Clinical research studies sponsored by AbbVie are subject to the International Council for Harmonisation (ICH) Good Clinical Practices (GCP) and local regulations and guidelines governing the study at the site location. In signing the Investigator Agreement, the investigator is agreeing to the following:

- 1. Conducting the study in accordance with ICH GCP, the applicable regulatory requirements, current protocol and operations manual, and making changes to a protocol only after notifying AbbVie and the appropriate Institutional Review Board (IRB)/Independent Ethics Committee (IEC), except when necessary to protect the subject from immediate harm.
- 2. Personally conducting or supervising the described investigation(s).
- 3. Informing all subjects, or persons used as controls, that the drugs are being used for investigational purposes and complying with the requirements relating to informed consent and ethics committees (e.g., IEC or IRB) review and approval of the protocol and its amendments.
- 4. Reporting complaints that occur in the course of the investigation(s) to AbbVie.
- 5. Reading the information in the Investigator's Brochure/safety material provided, including the instructions for use and the potential risks and side effects of the investigational product(s).
- 6. Informing all associates, colleagues, and employees assisting in the conduct of the study about their obligations in meeting the above commitments.
- 7. Maintaining adequate and accurate records of the conduct of the study, making those records available for inspection by representatives of AbbVie and/or the appropriate regulatory agency, and retaining all study-related documents until notification from AbbVie.
- 8. Maintaining records demonstrating that an ethics committee reviewed and approved the initial clinical protocol and all of its amendments.
- 9. Reporting promptly, all changes in the research activity and all unanticipated problems involving risks to human subjects or others, to the appropriate individuals (e.g., coordinating investigator, institution director) and/or directly to the ethics committees and AbbVie.
- 10. Providing direct access to source data documents for study-related monitoring, audits, IEC/IRB review, and regulatory inspection(s).

| | <u> </u> |
|---------------------------------------------------|----------|
| Signature of Principal Investigator | Date |
| Name of Driverical Investigator (eviated outsmed) | |
| Name of Principal Investigator (printed or typed) | |



# **APPENDIX C. LIST OF PROTOCOL SIGNATORIES**

| Name | Title | Functional Area |
|------|-------|-------------------------------|
| | | Clinical Program Development |
| | | Clinical Program Development |
| | | Medical Writing |
| | | Immunology Development |
| | | Data and Statistical Sciences |
| | | Data and Statistical Sciences |
| | | Clinical Pharmacology |



# APPENDIX D. ADDITIONAL ENDPOINT/ASSESSMENT DEFINITIONS

### Physician's Global Assessment of Disease Activity

Physician's Global Assessment of Disease Activity (visual analogue scale [VAS]) allows physicians to score on a 100 mm horizontal scale (0 being very low and 100 being very high) to assess the patient's current disease activity.

#### DAS28

The DAS is a combined index used to measure the disease activity in patients with RA. The DAS provides a score (between 0 and 10) indicating how active the disease is at the time of measurement. The calculation of the DAS28 score used either ESR or CRP.

The calculation of the DAS28 score will use ESR based on the following formula:

The calculation of the DAS28 score will use CRP based on the following formula:

PtGA represents patient's global assessment of disease activity; ESR is measured in mm/h, CRP is measured in mg/L, TJC28 and SJC28 represent total TJC and total SJC, respectively, based on the 28 joints (including the left and right side of the body).

American College of Rheumatology 20/50/70 Response (ACR20/50/70)

ACR20/50/70 is defined as

- At least 20%/50%/70% improvement in SJC compared to BL AND
- At least 20%/50%/70% improvement in TJC compared to BL AND
- At least 20%/50%/70% improvement in at least 3 out of the following 5 variables
  - 1. Patient's Assessment of RA Pain Intensity VAS
  - 2. Patient's Global Assessment of Disease VAS
  - 3. Physician's Global Assessment of Disease Activity VAS
  - 4. Patient's Assessment of Disability on HAQ-DI
  - 5. Serum high-sensitivity C-reactive protein (hs-CRP).

#### Clinical Disease Activity Index (CDAI)

The CDAI is a composite index for assessing disease activity based on the summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on visual analogue scale (VAS) (0 - 10 cm) for estimating disease activity. It has range from 0 to 76.



| Simplified Disease A | ctivity In | ıdex ( | SDAI |
|----------------------|------------|--------|------|
|----------------------|------------|--------|------|

The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity (VAS 0 - 10 cm) and level of CRP (mg/dl, normal < 1 mg/dl). It has a range from 0 to 86.



## APPENDIX E. JOINT EVALUATION WORKSHEET EXAMPLE

| | | | Subje | ct Rig | ht | | | | Subje | ct Lef | ft | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 0 = Abs<br>1 = Pre | | | NA: | placed<br>= No<br>sment | | 0 = Abs<br>1 = Pres | | | NA: | placed<br>= No<br>sment |
| JOINT<br>(Tick Correct Answer) | | in/<br>erness | Swe | lling | Jo | int | _ | in/<br>erness | Swe | lling | Jo | int |
| 1. Shoulder | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 2. Elbow | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 3. Wrist | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 4. Metacarpophalangeal I | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 5. Metacarpophalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 6. Metacarpophalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 7. Metacarpophalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 8. Metacarpophalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 9. Thumb Interphalangeal | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 10. Prox. Interphalangeal II | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 11. Prox. Interphalangeal III | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 12. Prox. Interphalangeal IV | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 13. Prox. Interphalangeal V | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| 14. Knee | 0 | 1 | 0 | 1 | 9 | NA | 0 | 1 | 0 | 1 | 9 | NA |
| TOTAL Joint Count | | | | | | | | | | | | |



# APPENDIX F. REPORTED OUTCOMES VAS



# APPENDIX G. HEALTH ASSESSMENT QUESTIONNAIRE DISABILITY INDEX







# APPENDIX I. RHEUMATOLOGY COMMON TOXICITY CRITERIA V.2.0

For designation of AE terms not shown in the Rheumatology Common Toxicity Criteria v.2.0 table, the approach described in the header row should be used.

### Rheumatology Common Toxicity Criteria v.2.0

Based on Woodworth TG, et al. Standardizing assessment of adverse effects in rheumatology clinical trials II. Status of OMERACT Drug Safety Working Group May 2006: OMERACT 8. Standardizing Assessment and Reporting of Adverse Effects in Rheumatology Clinical Trials: Enabling Description of Comparative Safety Profiles for Anti-Rheumatic Therapies.



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| A. Allergic/Immunologic | ic | | | |
| A1. Allergic reaction/<br>hypersensitivity<br>(includes drug fever) | Transient rash: drug fever < 38°C:<br>transient, asymptomatic<br>bronchospasm | Generalised urticaria responsive to<br>meds; or drug fever > 38°C, or<br>reversible bronchospasm | Symptomatic bronchospasm requiring meds; symptomatic urticaria persisting with meds, allergy related oedema/angioedema | Anaphylaxis, laryngeal/pharyngeal<br>oedema, requiring resuscitation |
| A2. Autoimmune<br>reaction | Seriologic or other evidence of autoimmune reaction, but patient asymptomatic: all organ function normal and no treatment is required (e.g., vitiligo) | Evidence of autoimmune reaction involving a non-essential organ or functions, requiring treatment other than immunosuppressive drugs (e.g., hypothyroidism) | Reversible autoimmune reaction involving function of a major organ or toxicity requiring short term immunosuppressive treatment (e.g., transient colitis or anaemia) | Causes major organ dysfunction, or progressive, not reversible, or requires long term administration of high dose immunosuppressive therapy |
| A3. Rhinitis (includes sneezing, nasal stuffiness, post nasal discharge) | Transient, non-prescription meds<br>relieve | Prescription meds required, slow | Corticosteroids or other prescription med with persistent disabling symptoms such as impaired exercise tolerance | NA |
| A4. Serum sickness | Transient, non-prescription meds<br>relieve | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Prolonged; symptoms only partially relieved by meds; parenteral corticosteroids required | Major organ dysfunction, requires<br>long-term high-dose<br>immunosuppressive therapy |
| A5. Vasculitis | Localised, not requiring treatment;<br>or rapid response to meds;<br>cutaneous | Symptomatic, slow response to meds (e.g., oral corticosteroids) | Generalised, parenteral corticosteroids required or/and short duration hospitalisation | Prolonged, hospitalisation, ischemic<br>changes, amputation |



| | <ul> <li>1 – Mild</li> <li>No medication or OTC</li> <li>Asymptomatic, or transient</li> <li>Short duration (&lt; 1 week)</li> <li>No change in life style</li> </ul> | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| B. Cardiac | | | | |
| B1. Arrhythmia | Transient, asymptomatic | Transient, but symptomatic or recurrent, responds to meds | Recurrent/persistent; maintenance prescription | Unstable, hospitalisation required, parenteral meds |
| B2. Cardiac function<br>decreased | Asymptomatic decline in resting ejection fraction by > 10%, but < 20% of baseline value | Asymptomatic decline of resting ejection fraction ≥ 20% of baseline value | CHF responsive to treatment | Severe or refractory CHF |
| B3. Edema | Asymptomatic (e.g., 1 + feet/calves), self-limited, no therapy required | Symptomatic (e.g., 2 + feet/calves), requires therapy | Symptoms limiting function (e.g., 3 + feet/calves, 2 + thighs), partial relief with treatment prolonged | Anasarca; no response to treatment |
| B4. Hypertension<br>(new onset or<br>worsening) | Asymptomatic, transient increase by > 20 mmHg (diastolic) or to > 150/100 if previously normal, no therapy required | Recurrent or persistent increase > 150/100 or by > 10 mmHg (diastolic), requiring and responding readily to treatment | Symptomatic increase > 150/100, > 20 mmHg, persistent, requiring multi agency therapy, difficult to control | Hypertensive crisis |
| B5. Hypotension<br>(without underlying<br>diagnosis) | Transient, intermittent, asymptomatic, orthostatic decrease in blood pressure > 20 mmHg | Symptomatic, without interference with function, recurrent or persistent > 20 mmHg decrease, responds to treatment | Syncope or symptomatic, interferes with function, requiring therapy and sustained medical attention, dose adjustment or drug discontinuation | Shock |
| B6. Myocardial<br>ischaemia | Transient chest pain/ECG changes;<br>rapid relief with nitro | Recurring chest pain, transient<br>ECG ST-T changes; treatment<br>relieves | Angina with infarction, no or<br>minimal functional compromise,<br>reduce dose or discontinue study<br>drug | Acute myocardial infarction,<br>arrhythmia or/and CHF |
| B7. Pericarditis/<br>pericardial effusion | Rub heard, asymptomatic | Detectable effusion by<br>echocardiogram, symptomatic<br>NSAID required | Detectable on chest x-ray, dyspnoea;<br>or pericardiocentesis; requires<br>corticosteroids | Pulsus alternates with low cardiac<br>output; requires surgery |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| B. Cardiac (continued) | | | | |
| B8. Phlebitis/thrombosis/ Embolism (excludes injection sites) | Asymptomatic, superficial,<br>transient, local, or no treatment<br>required | Symptomatic, recurrent, deep vein thrombosis, no anticoagulant therapy required | Deep vein thrombosis requiring anticoagulant therapy | Pulmonary embolism |
| C. General (Constitutional) | nal) | | | |
| C1. Fatigue/malaise<br>(asthenia) | Increase over baseline; most usual daily functions maintained, short term | Limits daily function intermittently over time | Interferes with basic ADL, persistent | Unable to care for self, bed or<br>wheelchair bound > 50% of day<br>debilitating, hospitalisation |
| C2. Fever (pyrexia)<br>(note: fever due to<br>drug allergy should be<br>coded as allergy) | Transient, few symptoms<br>37.7 – 38.5°C | Symptomatic, recurrent<br>38.6 – 39.9°C. Relieved by meds | ≥ 40°C; ≤ 24 h, persistent symptoms; partial response to meds. | > 40°C, debilitating, > 24 h,<br>hospitalisation; no relief with meds |
| C3. Headache | Transient or intermittent, no meds or relieved with OTC | Persistent, recurring, non-narcotic analgesics relieve | Prolonged with limited response to narcotic medicine | Intractable, debilitating, requires<br>parenteral meds. |
| C4. Insomnia | Difficulty sleeping, short term, no interfering with function | Difficulty sleeping interfering with function, use of prescription med. | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no<br>relief with meds |
| C5. Rigors, chills | Asymptomatic, transient, no meds, or non-narcotic meds relieve | Symptomatic, narcotic meds relieve. | Prolonged symptoms, with limited response to narcotic meds | Debilitating, hospitalisation; no relief with meds |
| C6. Sweating<br>(diaphoresis) | Episodic, transient | Frequent, short term | Frequent, drenching, disabling | Dehydration, requiring IV<br>fluids/hospitalization > 24 hrs |
| C7. Weight gain | 2% – 9.9% | 10% – 19.9% | 20% – 30% | NA |
| C8. Weight loss | 2% – 9.9% | 10% – 19.9% | 20% – 30% | NA |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| D. Dermatologic | | | | |
| D1. Alopecia | Subjective, transient | Objective, fully reversible | Patchy, wig used, partly reversible | Complete, or irreversible even if patchy |
| D2. Bullous eruption | Localised, asymptomatic | Localised, symptomatic, requiring treatment | Generalised, responsive to treatment; reversible | Prolonged, generalised, or requiring hospitalisation for treatment |
| D3. Dry skin | Asymptomatic, controlled with<br>emollients | Symptoms eventually (1 – 2 wks) controlled with emollients | Generalised, interfering with ADL<br>> 2 wks, persistent pruritis, partially<br>responsive to treatment | Disabling for extended period,<br>unresponsive to ancillary therapy<br>and requiring study drug<br>discontinuation for relief |
| D4. Injection site<br>reaction | Local erythema, pain, pruritis,<br>< few days | Erythema, pain, oedema, may<br>include superficial phlebitis,<br>1 – 2 wks | Prolonged induration, superficial<br>ulceration; includes thrombosis | Major ulceration necrosis requiring surgery |
| D5. Petechiae<br>(without vasculitis) | Few, transient asymptomatic | Dependent areas, persistent up to 2 wks | Generalised, responsive to treatment; reversible | Prolonged, irreversible, disabling |
| D6. Photosensitivity | Transient erythema | Painful erythema and oedema<br>requiring topical treatment | Blistering or desquamation, requires systematic corticosteroids | Generalised exfoliation or<br>hospitalisation |
| D7. Pruritis | Localised, asymptomatic, transient, local treatment | Intense, or generalised, relieved<br>by systematic medication | Intense or generalised; poorly<br>controlled despite treatment | Disabling, irreversible |
| D8. Rash (not<br>bullous) | Erythema, scattered<br>macular/popular eruption; pruritis<br>transient; TOC or no meds | Diffuse macular/popular eruption<br>or erythema with pruritus; dry<br>desquamation; treatment<br>required | Generalised, moist desquamation, requires systemic corticosteroids, responsive to treatment; reversible | Exfoliative or ulcerating; or requires hospitalisation; or parenteral corticosteroids |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| D. Dermatologic (continued) | nued) | | | |
| D9. Induration/<br>fibrosis/Thickening<br>(not sclerodermal) | Localized, high density on<br>palpation, reversible, no effect on<br>ADL and not disfiguring | Local areas < 50% body surface,<br>not disfiguring, transient<br>interference with ADL, reversible | Generalized, disfiguring, interferes<br>with ADL, reversible | Disabling, irreversible, systemic<br>symptoms |
| E. Ear/Nose/Throat | | | | |
| E1. Hearing loss | Transient, intermittent, no interference with function | Symptomatic, treatment required, reversible | Interferes with function; incomplete response to treatment | Irreversible deafness |
| E2. Sense of smell | Slightly altered | Markedly altered | Complete loss, reversible | Complete loss, without recovery |
| E3. Stomatitis | Asymptomatic | Painful, multiple, can eat | Interferes with nutrition, slowly reversible | Requires enteral support; residual dysfunction |
| E4. Taste disturbance<br>(dysgeusia) | Transiently altered; metallic | Persistently altered; limited effect on eating | Disabling, effect on nutrition | NA |
| E5. Tinnitus | Intermittent, transient, no<br>interference with function | Requires treatment, reversible | Disabling, or associated with hearing loss | Irreversible deafness |
| E6. Voice changes<br>(includes hoarseness,<br>loss of voice, laryngitis) | Intermittent hoarseness, able to<br>vocalise | Persistent hoarseness, able to vocalise | Whispered speech, slow return of ability to vocalise | Unable to vocalize for extended |
| E7. Xerostomia (dry<br>mouth) | Transient dryness | Relief with meds | Interferes with nutrition, slowly reversible | Extended duration interference with nutrition, requires parenteral nutrition |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| F. Eye/Ophthalmologic | | | | |
| F1. Cataract | Asymptomatic, no change in vision,<br>non-progressive | Symptomatic, partial visual loss,<br>progressive | Symptoms impairing function, vision loss requiring treatment, including surgery | NA |
| F2. Conjunctivitis | Asymptomatic, transient, rapid<br>response to treatment | Symptomatic, responds to treatment, changes not interfering with function | Symptoms prolonged, partial response to treatment, interferes with function | NA |
| F3. Lacrimation<br>increased (tearing,<br>watery eyes) | Symptoms not requiring treatment, transient | Symptomatic, treatment required, reversible | Unresponsive to treatment with<br>major effect on function | NA |
| F4. Retinopathy | Asymptomatic, non-progressive, no<br>treatment | Reversible change in vision; readily responsive to treatment | Disabling change in vision ophthalmological findings reversible, sight improves over time | Loss of sight |
| F5. Vision changes<br>(e.g., blurred,<br>photophobia, night<br>blindness, vitreous<br>floaters) | Asymptomatic, transient, no<br>treatment required | Symptomatic, vision changes not interfering with function, reversible | Symptomatic, vision changes<br>interfering with function | Loss of sight |
| F6. Xerophtalmia (dry<br>eyes) | Mild scratchiness | Symptomatic without interfering with function, requires artificial tears | Interferes with vision/function,<br>corneal ulceration | Loss of sight |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| G. Gastrointestinal | | | | |
| G1. Anorexia | Adequate food intake, minimal<br>weight loss | Symptoms requiring oral nutritional supplementation | Prolonged, requiring iv support | Requires hospitalization for nutritional support |
| G2. Constipation | Asymptomatic, transient, responds to stool softener, OTC laxatives | Symptomatic, requiring prescription laxatives, reversible | Obstipation requiring medical intervention | Bowel obstruction. Surgery required. |
| G3. Diarrhea | Transient, increase of 2 – 3 stools/day over pretreatment (no blood or mucus), OTC agents relieve | Symptomatic, increase<br>4 – 6 stools/day, nocturnal stools,<br>cramping, requires treatment with<br>prescription meds. | Increase > 6 stools/day, associated with disabling symptoms, e.g., incontinence, severe cramping, partial response to treatment. | Prolonged, dehydration,<br>unresponsive to treatment,<br>requires hospitalization. |
| G4. Dyspepsia<br>(heartburn) | Transient, intermittent, responds<br>to OTC antacids, H-2 blockers | Prolonged, recurrent, requires<br>prescription meds, relieved by<br>meds | Persistent despite treatment,<br>interferes with function, associated<br>with GI bleeding | NA |
| G5. GI bleed<br>(gastritis, gastric or<br>duodenal ulcer<br>diagnosed-define<br>aetiology) | Asymptomatic, endoscopic finding, haemocult + stools, no transfusion, responds rapidly to treatment | Symptomatic, transfusion ≤ 2 units<br>needed; responds to treatment | Haematemesis, transfusion<br>3 – 4 units, prolonged interference<br>with function | Recurrent, transfusion > 4 units, perforation, requiring surgery, hospitalisation |
| G6. Haematochezia<br>(rectal bleeding) | Haemorrhodial, asymptomatic, no<br>transfusion | Symptomatic, transfusion<br>< 2 units, reversible | Recurrent, transfusion > 3 – 4 units | > 4 units, hypotension, requiring hospitalization |
| G7. Hepatitis | Laboratory abnormalities,<br>asymptomatic, reversible | Symptomatic laboratory abnormalities, not interfering with function, slowly reversible | Laboratory abnormalities persistent > 2 wks, symptoms interfere with function | Progressive, hepato-renal,<br>anasarca, pre-coma or coma |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| G. Gastrointestinal (continued) | ntinued) | | | |
| G8. Nausea, or<br>nausea/vomiting (use<br>diagnostic term) | Transient, intermittent, minimal interference with intake, rapid response to meds. | Persistent, recurrent, requires<br>prescription meds, intake<br>maintained | Prolonged, interferes with daily function and nutritional intake, periodic iv fluids | Hypotensive, hospitalization, parenteral nutrition, unresponsive to out-patient management |
| G9. Pancreatitis | Anylase elevation, intermittent<br>nausea/vomiting, transient,<br>responds rapidly to treatment | Amylase elevation with abdominal pain, nausea, occasional vomiting, responsive to treatment | Severe, persistent abdominal pain with pancreatitic enzyme elevation, incomplete or slow response to treatment | Complicated by shock,<br>haemorrhage (acute circulatory<br>failure) |
| G10. Proctitis | Perianal pruritus, haemorrhoids<br>(new onset), transient, or<br>intermittent, relieved by OTC meds | Tenesmus or ulcerations, anal fissure, responsive to treatment, minimal interference with function | Unresponsive to treatment, marked interference with function | Mucosal necrosis with<br>haemorrhage, infection, surgery<br>required. |
| H. Musculoskeletal | | | | |
| H1. Avascular<br>necrosis | Asymptomatic MRI changes, non-<br>progressive | MRI changes and symptoms responsive to rest and analgesia | MRI changes, symptoms requiring surgical intervention | Wheelchair bound; surgical repair not possible |
| H2. Arthralgia | Intermittent transient symptoms,<br>no meds or relieved by OTC meds | Persistent or recurrent symptoms, resolve with meds, little effect on function | Severe symptoms despite meds<br>impairs function | Debilitating, hospitalisation<br>required for treatment |
| H3. Leg cramps | Transient, intermittent, does not interfere with function | Recurrent symptoms, minimally interferes with function or sleep, responds to meds | Persistent, prolonged interference<br>with function or sleep, partial or no<br>response to meds | NA |
| H4. Myalgia | Occasional; does not interfere with function | Frequent, requires meds (non-<br>narcotic); minor effects on<br>function | Major change in function/lifestyle,<br>narcotic pain meds | Debilitating, profound weakness, requires wheelchair, unresponsive to meds |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| I. Neuropsychiatric | | | | |
| <ol> <li>Anxiety or<br/>Depression (mood<br/>alteration)</li> </ol> | Symptomatic, does not interfere with function; no meds | Frequent symptoms, responds to<br>meds; interferes with ADL at times | Persistent, prolonged symptoms, partial or no response to meds, limits daily function | Suicidal ideation or danger to self |
| <ol> <li>Cerebrovascular ischaemia</li> </ol> | NA | Single transient ischaemic event, responsive to treatment | Recurrent transient ischaemic<br>events | Cerebrovascular vascular accident with permanent disability |
| 13. Cognitive<br>disturbance | Subjective symptoms, transient, intermittent, not interfering with function | Objective symptoms, persisting, interferes with daily function occasionally | Persistent, or worsening objective symptoms; interferes with routine daily routine | Debilitating/disabling and permanent; toxic psychosis |
| <ul><li>14. Depressed consciousness</li><li>(somnolence)</li></ul> | Observed, transient, intermittent,<br>not interfering with function | Somnolence or sedation,<br>interfering with function | Persistent, progressive, obundation, stupor | Coma |
| <ol> <li>Inability to concentrate</li> </ol> | Subjective symptoms, does not interfere with function | Objective findings, interferes with function | Persistent, prolonged objective findings or organic cause | NA |
| 16. Insomnia (in<br>absence of pain) | Occasional difficulty sleeping,<br>transient intermittent, not<br>interfering with function | Recurrent difficulty sleeping; requires meds for relief; occasional interference with function | Persistent or worsening difficulty sleeping; severely interferes with routine daily function | NA |
| I7. Libido decreased | Decrease in interest | Loss of interest; influences<br>relationship | Persistent, prolonged interfering with relationship | NA |
| I8. Peripheral motor<br>neuropathy | Subjective or transient loss of deep tendon reflexes; function maintained | Objective weakness, persistent, no significant impairment of daily function | Objective weakness with substantial impairment of function | Paralysis |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| I. Neuropsychiatric (continued) | ntinued) | | | |
| <ul><li>19. Peripheral sensory neuropathy (sensory disturbance)</li></ul> | Subjective symptoms without objective findings, transient, not interfering with function | Objective sensory loss, persistent,<br>not interfering with function | Prolonged sensory loss or<br>paraethesias interfering with<br>function | NA |
| l10. Seizure | NA | Recurrence of old seizures,<br>controlled with adjustment of<br>meds | Recurrence/exacerbation with partial response to medication | Recurrence not controlled,<br>requiring hospitalization; new<br>seizures |
| I11. Vertigo<br>(dizziness) | Subjective symptoms, transient, intermittent, no treatment | Objective findings, recurrent,<br>meds relieve, occasionally<br>interfering with function | Persistent, prolonged, interfering with daily function; partial response to medication | Debilitating without response to<br>medication, hospitalization |
| J. Pulmonary | | | | |
| J1. Asthma | Occasional wheeze, no interference<br>with activities | Wheezing, requires oral meds, occasional interference with function | Debilitating, requires nasal O <sub>2</sub> | Requires ventilator assistance |
| J2. Cough | Transient, intermittent, occasional<br>OTC meds relieve | Persistent, requires narcotic or<br>other prescription meds for relief | Recurrent, persistent coughing spasms without consistent relief by meds, interferes with function | Interferes with oxygenation;<br>debilitating |
| J3. Dyspnea | Subjective, transient, no<br>interference with function | Symptomatic, intermittent or<br>recurring, interferes with<br>exertional activities | Symptomatic during daily routine activities, interferes with function, treatment with intermittent nasal O <sub>2</sub> relieves | Symptomatic at rest, debilitating,<br>requires constant nasal O <sub>2</sub> |
| J4. Pleuritic pain<br>(pleurisy) | Transient, intermittent symptoms,<br>no treatment or OTC meds relieve | Persistent symptoms, requires<br>prescription meds for relief | Prolonged symptoms, interferes<br>with function, requires frequent<br>narcotic pain relief | Debilitation, requiring<br>hospitalisation |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| J. Pulmonary (continued) | (p: | | | |
| J5. Pneumonitis<br>(pulmonary<br>infiltrates) | Asymptomatic radiographic changes, transient, no treatment required | Symptomatic, persistent, requiring corticosteroids | Symptomatic, requiring treatment including O <sub>2</sub> | Debilitating, not reversible; or requiring assisted ventilation |
| J6. Pulmonary<br>function decreased<br>(FVC or carbon<br>monoxide diffusion<br>capacity – DLCO) | 76% – 90% of pre-treatment value | 51% – 75% of pre-treatment value | 26% – 50% of pre-treatment value | < 25% of pre-treatment value |
| Laboratory Data | | | | |
| K. Haematology | | | | |
| K1. Hgb (g/dl)<br>decrease from pre-<br>treatment | 1.0 – 1.4 | 1.5-2.0 | 2.1 – 2.9, or Hgb < 8.0, > 7.0 | ≥ 3.0; or Hgb < 7.0 |
| K2. Leukopenia (total<br>WBC) × 1000 | 3.0 – 3.9 | 2.0-2.9 | 1.0 – 1.9 | < 1.0 |
| K3. Neutropenia<br>(× 1000) | 1.5 – 1.9 | 1.0-1.4 | 0.5 – 0.9 | < 0.5 |
| K4. Lymphopenia<br>(× 1000) | 1.5 – 1.9 | 1.0 – 1.4 | 0.5 – 0.9 | < 0.5 |
| K5. Platelets (× 1000) | 75 – LLN | 50 – 74.9 | 20 – 49.9; platelet transfusion required | < 20; recurrent platelet transfusions |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| L. Chemistry | | | | |
| L1. Hypercalcaemia<br>(mg/dl) | 1.1 × ULN – 11.5 | 11.6 – 12.5 | 12.6 – 13.5; or symptoms present | > 13.5; or associated coma |
| L2. Hyperglycemia<br>(mg/dl) Fasting | 140 – 160 | 161 – 250 | 251-500 | > 500, or associated with<br>ketoacidosis |
| L3. Hyperkalaemia<br>(mg/dl) | 5.5 – 5.9 | 6.0 – 6.4 | 6.5 – 7.0 or any ECG change | > 7.0 or any arrhythmia |
| L5. Hypocalcaemia<br>(mg/dl) | 0.9 × LLN – 7.8 | 7.7 – 7.0 | 6.9 – 6.5; or associated with symptoms | < 6.5 or occurrence of tetany |
| L6. Hypoglycemia<br>(mg/dl) | 55 – 64 (no symptoms) | 40 – 54 (or symptoms present) | 30 – 39 (symptoms impair function) | < 30 or coma |
| L7. Hyponatraemia<br>(mg/dl) | - | 125 – 129 | 120 – 124 | < 120 |
| L8. Hypokalaemia<br>(mg/dl) | - | 3.0 – 3.4 | 2.5 – 2.9 | < 2.5 |
| L9. CPK (also if polymyositis-disease) | 1.2 – 1.9 × ULN | 2.0-4.0×ULN | 4.0 × ULN with weakness but without life-threatening signs or symptoms | > 4.0 × ULN with signs or symptoms of rhabdomyolysis or life-threatening |
| L10. Serum uric acid | $1.2 - 1.6 \times ULN$ | 1.7 – 2.9 × ULN | 3.0 – 5.0 × ULN or gout | NA |
| L11. Creatinine<br>(mg/dL) | 1.1 – 1.3 × ULN | 1.3 – 1.8 × ULN | 1.9 – 3.0 × ULN | > 3.0 × ULN |
| L12. SGOT (AST) | 1.2 – 1.5 × ULN | 1.6 – 3.0 × ULN | 3.1 – 8.0 × ULN | > 8.0 × ULN |
| L13. SGPT (ALT) | 1.2 – 1.5 × ULN | 1.6-3.0 × ULN | 3.0 – 8.0 × ULN | > 8.0 × ULN |



| | 1 – Mild No medication or OTC Asymptomatic, or transient Short duration (< 1 week) No change in life style | 2 – Moderate Symptomatic Duration (1 – 2 weeks) Alter lifestyle occasionally Meds relieve (may be prescription) Study drug continued | 3 – Severe Prolonged symptoms, reversible, major functional impairment Prescription meds/partial relief May be hospitalized < 24 hr Temporary study drug discontinuation or/and dose reduced | 4 – Includes Life Threatening At risk of death Substantial disability, especially if permanent Multiple meds Hospitalized > 24 hr Study drug discontinued |
|---|---|---|---|---|
| L. Chemistry (continued) | (p: | | | |
| L14. Alkaline<br>phosphatase | 1.1 – 2.0 × ULN | 1.6 – 3.0 × ULN | 3.0 – 5.0 × ULN | > 5.0 × ULN |
| L15. T. bilirubin | 1.1 – 1.4 × ULN | 1.5 – 1.9 × ULN | 2.0 – 3.0 × ULN | > 3.0 × ULN |
| L16. LDH | $1.3 - 2.4 \times ULN$ | 2.5 – 5.0 × ULN | 5.1 – 10 × ULN | > 10 × ULN |
| M. Urinalysis | | | | |
| M1. Haematuria | Micro only | Gross, no clots | Clots, transfusion < 2 units | Transfusion required |
| M2. Proteinuria (per<br>24 h) | 300 – 500 mg (tr/1+) | 501 – 1999 mg (2+) | 2 – 5.0 g (3+) nephrotic syndrome | 5.0 g (4+) anasarca |
| M3. WBC in urine | NA | NA | Indicating acute interstitial nephritis | Associated with acute renal failure |
| M4. Uric acid crystals | Present without symptoms | NA | With stones or symptoms of stones (e.g., renal colic) | Causing renal outflow obstruction and hospitalization |

ADL = activities of daily living; ANA = antinuclear antibodies; CHF = congestive heart failure; ECG = electrocardiogram; FVC = forced vital capacity; H-2 blockers = histamine-2 blockers IV = intravenous; LLN = lower limit of normal; MRI = magnetic resonance imaging; OTC = over-the-counter medication; SLE = systemic lupus erythematosus; ULN = upper limit of normal; WBC = white blood cells



# APPENDIX J. ACTIVITY SCHEDULE

The following table shows the required activities the subject encounters. The individual activities are described in detail in Appendix K, the **Operations Manual**.

# abbvie

Study Activities Table

| | Screening | Baseline | u t | 2 Wk | W 4 | e Wk | % Wk | 10 Wk | 0<br>72 | D 0 73 | 11 Wk | 12 W | 14 WK | wk 16 | 18 V | 20 Wk | 75 WK | 74 Wk | Premature<br>Discontinuation | 70-Day F/U<br>contact |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | Day –35 to<br>Day 1 | I yed | 8 yed | SI yed | 62 yed | Day 43 | 72 ysQ | L7 yed | 27 ysd | £7 ysQ | 87 yed | Z8 yed | 66 YeQ | Day 113 | TS1 yed | Day 141 | Day 155 | 691 YEQ | | |
| ☐ INTERVIEWS & QUESTIONNAIRES | IRES | | | | | | | | | | | | | | | | | | | |
| Subject information and informed consent | > | | | | | | | | | | | | | | | | | | | |
| Eligibility criteria | 8 | > | | | | | | | | | | | | | | | | | | |
| Medical/surgical history | * | 1 | | | | | | | | | | | | | | | | | | |
| Alcohol and nicotine use | * | | | | | | | | | | | | | | | | | | | |
| Adverse event assessment | > | * | × | \$ | Ş | × | <b>S</b> | \$ | | | | <b>S</b> | > | > | \$ | <u> </u> | <b>y</b> | \$ | Ş | ¥ |
| Prior/concomitant therapy | * | * | × | × | Ş | ¥ | > | S. | | | | • | > | * | * | <b>\$</b> | , | * | * | * |
| Latent TB risk assessment form | V | | 80 | | | | | | | | | | | - 6 | | 8 | | | 50 | |
| Patient's Assessment of Pain | À | À | > | × | × | × | × | Ş | | 8 | | > | | > | \$ | ×. | * | Ş | > | |
| Patient's Assessment of Disease Activity | > | \$ | > | > | > | > | ` | > | | - 85 | | \$ | ` | > | ` | <b>\</b> | \$ | \$ | > | |
| HAQ-DI | | À | × | À | > | × | > | > | | 25 | | | | 9 | | <u> </u> | Ş | | > | |
| SF-36 | | \$ | (): | 00 | | | | | | | | > | | 09<br>09 | <i>i</i> | ()<br>() | | × | * | |
| 👚 LOCAL LABS & EXAMS | | | | | | | | | | | | | | | | | | | | |
| Body Weight | * | > | | | | | | | | | | > | | | | | | | | |
| Height | J. | | | | | | | | | | | | | a de | | i i | | | | |
| Vital Signs <sup>a</sup> | * | \$ | × | \$ | > | × | > | \$ | | | | <b>&gt;</b> | | 8 | | \$ | | \$ | ~ | |
| Physical Exam | 8 | > | | | | | | | | | | \$ | | | $\vdash$ | | | 8 | * | |

STUDY M16-560 | Version 5.0 | EudraCT 2018-003053-21 CONFIDENTIAL INFORMATION No use or disclosure outside AbbVie is permitted without prior written authorization from AbbVie.

# abbvie

| | Screening | Baseline | 1 Wk | 2 Wk | Wk 4 | w e | wk 1 | Wk 10 1 | D 27 | V D V | Wk W | Wk W | Wk v | Wk Wk<br>16 18 | k Wk | k Wk | k Wk | Premature<br>Discontinuation | U/1 YEG-07 | contact |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Activity | Day –35 to | T yed | Day 8 | Day 15 | 62 yed | EA YEG | 72 yed | IT yed | 27 yed | ET yed | 87 Yed | 28 Yea | 66 Yed | Day 113 | TSI YEG | Day 141 | 697 Yed | | | |
| 12-lead ECG | > | | | | | .9 8 | 9 8 | | | 8 8 | | > | | 2 | | 2 6 | > | > | | |
| Chest x-ray | > | | | | | .9 | 9 | | | 8 | Si. | | | 3 | | 2 | | | | |
| ESR | | \$ | × | \$ | > | > | × | > | | | | \$ | Š | <i>&gt;</i> | > | · | > | > | | |
| Physician's Global Assessment of Disease<br>Activity | 5 | 5 | ~ | - 18 | > | ~ | × | 8 | | | | , | , · | , | * | • | 3 | * | | |
| TJC28 and SJC28 | \$ | ` | × | <b>S</b> | > | <b>×</b> | <b>×</b> | 8 | | | | · . | | 1 | * | <b>&gt;</b> | * | <b>&gt;</b> | | |
| Urine pregnancy test (for all female subjects of childbearing age) | | <b>\$</b> | | | \$ | | <b>S</b> | | | | | <b>\</b> | 343 | S | > | | • | * | | |
| TCENTRAL LABS | | ā S | | 9 | | š : | 9 | ā ā | 6 1 | e a | <u> </u> | 8 | ā 8 | [ | 9 | | <b>3</b> | 5 | <b>G</b> 9 | |
| Serum pregnancy test (for all female subjects of childbearing age) | <b>&gt;</b> | | | | | | | | | | | | | | | | | | | |
| hsCRP | 5 | > | ¥ | > | * | ¥ | × | > | | | | S . | · · | 1 | > | <i>*</i> | A | A | | |
| Hematology <sup>b</sup> | * | ` | > | > | > | * | ` | | | | | > | , V | > | • | | 7 | <b>*</b> | | |
| Clinical chemistry and urinalysis | > | \$ | | > | ¥ | | > | | | 8 | | 1 | 26 | ~ | > | | > | × | | |
| TB Test (QuantiFERON TB Gold test and/or local purified protein derivative (tuberculin) skin test, if required) | S | | S 80 | | | | 9 | | | 8 | %) = ================================== | | | 20 E | | 3 S | | | | |
| HIV, HAV, HBV, and HCV | > | | | | | 9.5 | 9 | | | 8 | 62 | | | | | | | | | |
| Blood samples for conjugated ADC<br>ABBV-3373 (serum), total antibody (serum),<br>free A-1677770 (plasma) assays, and<br>adalimumab assays <sup>c</sup> | | \$ | > | <b>S</b> | J. J. | <b>&gt;</b> | | <b>\$</b> | | | | \$ | , | | >= | | · · | ` | | |

STUDY M16-560 | Version 5.0 | EudraCT 2018-003053-21 CONFIDENTIAL INFORMATION No use or disclosure outside AbbVie is permitted without prior written authorization from AbbVie.



| 691 Aed | gninseroc | Baseline | 1 W | Wk WI | | % % | 8 Wk | 10 T | D D 72 73 | 11 W | 12 W. | W. 41 | Wk<br>16 | WK<br>18 | Wk<br>20 | Wk<br>22 | Wk<br>24 | Premature<br>Discontinuation | U\P Y0-Day F\U<br>contact |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day –35 to | T yed | 8 yed | 92 | | SAME STATE | | | | Made and | o entre approprie | | Day 113 | TSI YEG | Day 141 | Day 155 | 691 Yed | | |
| | | \$ | 3 | | | 87 | 9 | | | 8 | 1 | | | | a a | | * | * | |
| | | > | S | | | | | | | | > | | > | | | | | | |
| | 1 8 | | | | | - P | S 62 | | | | 7 13 | > | | | | | | | |
| | <u> </u> | <b>S</b> | <b>\</b> | 8 | | 12 | | | | ж | > | | 8 | | * | | À | * | |
| | <del>-</del> | - 5 | × . | × . | | | | | | | - > | | * | 10 | × . | | de la constantina | * | |
| | | \$ | > | 8 | 163 | | | | | | \$ | | 88 | | | | \$ | * | |
| | | > | × | ¥ | * | ~ | | | | | > | | × | | | | 1 | 1 | |
| | | 5 | | | | | | | | | | | | | | | | | |
| | | | | | | | | | ŝ | | | | | | | | | | |
| | V. | \$ | | | | - 50 | 67 | | | - 8 | - | | | | | | | | |
| | | \$ | 1 1 | -22<br> | | | | <u> </u> | | 8 8 | > | > | × | ۶ | > | Ş | | | |

| Administration study drug/placebo | | | | > | > | > | > | > | | 8 8 | | \$<br>*<br>\ | | > | \$ | Ц |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| oird parisseam of Ilim origana boold | rtos | nd 20 | min of | to Wet | and when | apr bi | niniotes | tion / | W oto | 100 | . otho | <br>- III. | a charle | 0.000 | ouc p | |

- blood pressure will be measured prior to and 30 min after IV study drug administration (up to Week 10); otherwise, it will only be measured once.
- HbA1c will be assessed at Screening, Week 12, and Week 24. þ.
- Pre-dose PK samples will be taken on dosing days. PK samples will also be taken at 1 hour and 3 hours after IV administration (from the contralateral arm) on Day 1 and Day 71. j
- Additional PK samples will be collected for subjects who consent to participating in the optional intensive PK sampling (D72, D73 and D78).



## APPENDIX K. SUMMARY OF CHANGES

#### **Previous Protocol Versions**

| Protocol | Date |
|------------------------------|------------------|
| Version 1.0 | 18 October 2018 |
| Version 1.1 (Germany Only) | 07 November 2019 |
| Version 1.1.1 (Germany Only) | 20 November 2019 |
| Version 2.0 | 20 November 2019 |
| Version 3.0 | 20 November 2019 |
| Version 4.0 | 11 March 2020 |
| Version 4.1 (Germany Only) | 12 March 2020 |

The purpose of this version is to remove the cohort. Minor clerical edits have been made as needed for consistency and clarity throughout the protocol.

## **Summary of Protocol Changes:**



Section 4.2, removed details of study conduct related to







| • | Section 1, added section description for clarity, and removed from Pharmacokinetic Lab section. |
|---|---|
| | Rationale: is not being studied in this protocol. |
| • | Section 2.1, removed study activities for the section 2.1. |
| | Rationale: is not being studied in this protocol. |
| • | Section 3.5, removed sections for PK and immunogenicity sampling for |
| | Rationale: is not being studied in this protocol. |
| • | Section 3.6, removed biomarker sampling for . |
| | Rationale: is not being studied in this protocol. |
| • | Section 3.12, removed clinical laboratory testing for the cohort. |
| | Rationale: is not being studied in this protocol. |
| • | Section 5.1, removed for SUSAR reporting. |
| | Rationale: is not being studied in this protocol. |
| • | Section 6.1, removed section for treatment administration. |
| | Rationale: is not being studied in this protocol. |
| • | Section 6.2, removed information on for drug supply, storage, and disposition. |
| | Rationale: is not being studied in this protocol. |
| • | Section 6.3, removed the section for method of assigning subjects to treatment groups for the cohort. |
| | Rationale: is not being studied in this protocol. |
| • | Section 6.4, removed the section for timing of study drug in the cohort. |
| | Rationale: is not being studied in this protocol. |



# APPENDIX L. OPERATIONS MANUAL